CLINICAL TRIAL: NCT00430521
Title: Reactogenicity and Immunogenicity Study of GlaxoSmithKline Biologicals' Pandemic Influenza Vaccine (GSK1119711A) Administered According to Different Vaccination Schedules
Brief Title: Safety & Immunogenicity of an Alternative Immunization Schedule of GSK Bio's Pandemic Influenza Vaccine (GSK1119711A)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 107495; 2006-005477-22 (EudraCT Number)
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Results first posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Influenza; Influenza Vaccines
Keywords: Pandemic Flu; Pandemic influenza vaccine (GSK1119711A)
MeSH Terms: conditions — Influenza, Human

ARMS (8):
- GSK1562902A V/I/6 Group (Experimental): Subjects received 1 dose of vaccine formulated from VT strain at Day 0 and 1 dose of the vaccine including IN at Month 6. The vaccine was administered in the deltoid region of the non-dominant arm.
  Interventions: Biological: Pandemic influenza vaccine (GSK1119711A)-formulation 1; Biological: Pandemic influenza vaccine (GSK1119711A)-formulation 2
- GSK1562902A V/V/6 Group (Experimental): Subjects received 2 doses of vaccine formulated from VT strain, 1 at Day 0 and 1 at Month 6. The vaccine was administered in the deltoid region of the non-dominant arm.
  Interventions: Biological: Pandemic influenza vaccine (GSK1119711A)-formulation 1
- GSK1562902A 2V/I/6 Group (Experimental): Subjects received 2 doses of vaccine formulated from VT strain, 1 at Day 0 and 1 at Day 21 and a 3rd dose of vaccine including IN strain at Month 6.The vaccine was administered in the deltoid region of the non-dominant arm.
  Interventions: Biological: Pandemic influenza vaccine (GSK1119711A)-formulation 1; Biological: Pandemic influenza vaccine (GSK1119711A)-formulation 2
- GSK1562902A 2V/V/6 Group (Experimental): Subjects received 2 doses of vaccine formulated from VT strain, 1 at Day 0 and 1 at Day 21 and a 3rd dose of vaccine including VT strain at Month 6. The vaccine was administered in the deltoid region of the non-dominant arm.
  Interventions: Biological: Pandemic influenza vaccine (GSK1119711A)-formulation 1
- GSK1562902A V/I/12 Group (Experimental): Subjects received 1 dose of vaccine formulated from VT strain at Day 0 and 1 dose of the vaccine including IN strain at Month 12. The vaccine was administered in the deltoid region of the non-dominant arm.
  Interventions: Biological: Pandemic influenza vaccine (GSK1119711A)-formulation 1; Biological: Pandemic influenza vaccine (GSK1119711A)-formulation 2
- GSK1562902A V/V/12 Group (Experimental): Subjects received 2 doses of vaccine formulated from VT strain, 1 at Day 0 and 1 at Month 12. The vaccine was administered in the deltoid region of the non-dominant arm.
  Interventions: Biological: Pandemic influenza vaccine (GSK1119711A)-formulation 1
- GSK1562902A 2V/I/12 Group (Experimental): Subjects received 2 doses of vaccine formulated from VT strain, 1 at Day 0 and 1 at Day 21 and a 3rd dose of vaccine including IN strain at Month 12.The vaccine was administered in the deltoid region of the non-dominant arm.
  Interventions: Biological: Pandemic influenza vaccine (GSK1119711A)-formulation 1; Biological: Pandemic influenza vaccine (GSK1119711A)-formulation 2
- GSK1562902A 2V/V/12 Group (Experimental): Subjects received 2 doses of vaccine formulated from VT strain, 1 at Day 0 and 1 at Day 21 and a 3rd dose of vaccine including VT strain at Month 12.The vaccine was administered in the deltoid region of the non-dominant arm.
  Interventions: Biological: Pandemic influenza vaccine (GSK1119711A)-formulation 1

INTERVENTIONS:
Biological: Pandemic influenza vaccine (GSK1119711A)-formulation 1 — 2 or 3 doses, intramuscular injection, at different time points.
  Other Names: VT strain
Biological: Pandemic influenza vaccine (GSK1119711A)-formulation 2 — 2 or 3 doses, intramuscular injection, at different time points.
  Other Names: IN strain
  Arms: GSK1562902A 2V/I/12 Group; GSK1562902A 2V/I/6 Group; GSK1562902A V/I/12 Group; GSK1562902A V/I/6 Group

SUMMARY:
The aim of the study is to assess the safety & immunogenicity of a pandemic influenza vaccine administered at 2 different time points. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female between, and including, 18 and 60 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* If the subject is female, she must be of non-childbearing potential; or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions for 30 days prior to first vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series.

Exclusion Criteria:

* Administration of licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrolment in this study.
* History of vaccination with investigational influenza pandemic vaccine.
* History of administration of an experimental/licensed vaccine
* Planned administration of a vaccine not foreseen by the study protocol during the following periods: from Day 0 up to Day 51; from 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to Month 6 and Month 12; from Month 6 up to Month 6 + 30 days; from Month 12 up to Month 12 + 30 days.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first administration of the candidate vaccines
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* History of hypersensitivity to vaccines.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* History of chronic alcohol consumption and/or drug abuse.
* Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Serious chronic disease including any medically significant chronic pulmonary, cardiovascular, renal, neurological, psychiatric or metabolic disorder, as determined by medical history and physical examination.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first administration of the candidate vaccine or during the study.
* Lactating women.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days prior to the first vaccination, or planned use during the study period.
* Any condition which, in the opinion of the investigator, prevents the subject from participation in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 512 (Actual)
Dates: Start 2007-02-05 (Actual); Primary Completion 2008-10-20 (Actual); Study Completion 2008-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- Germany (10):
  - GSK Investigational Site, Deggendorf, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Neu-Ulm, Bavaria
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Gillard P, Caplanusi A, Knuf M, Roman F, Walravens K, Moris P, Drame M, Schwarz TF. An assessment of prime-boost vaccination schedules with AS03A -adjuvanted prepandemic H5N1 vaccines: a randomized study in European adults. Influenza Other Respir Viruses. 2013 Jan;7(1):55-65. doi: 10.1111/j.1750-2659.2012.00349.x. Epub 2012 Mar 9. PMID 22405557
- [Background] Schwarz TF, Horacek T, Knuf M, Damman HG, Roman F, Drame M, Gillard P, Jilg W. Single dose vaccination with AS03-adjuvanted H5N1 vaccines in a randomized trial induces strong and broad immune responsiveness to booster vaccination in adults. Vaccine. 2009 Oct 23;27(45):6284-90. doi: 10.1016/j.vaccine.2009.01.040. PMID 19856521
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 107495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 107495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 107495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- GSK1562902A V/I/6 Group: Healthy male or female subjects, between and including 18 and 60 years of age, who received 1 dose of vaccine formulated from VT (A/Vietnam/1994/2004) strain at Day 0 and 1 dose of the vaccine including IN (A/Indonesia/05/2005) strain at Month 6. The vaccine was administered in the deltoid region of the non-dominant arm.
- GSK1562902A V/V/6 Group: Healthy male or female subjects, between and including 18 and 60 years of age, who received 2 doses of vaccine formulated from VT (A/Vietnam/1994/2004) strain, 1 at Day 0 and 1 at Month 6. The vaccine was administered in the deltoid region of the non-dominant arm.
- GSK1562902A 2V/I/6 Group: Healthy male or female subjects, between and including 18 and 60 years of age, who received 2 doses of vaccine formulated from VT (A/Vietnam/1994/2004) strain, 1 at Day 0 and 1 at Day 21 and a 3rd dose of vaccine including IN (A/Indonesia/05/2005) strain at Month 6.The vaccine was administered in the deltoid region of the non-dominant arm.
- GSK1562902A 2V/V/6 Group: Healthy male or female subjects, between and including 18 and 60 years of age, who received 2 doses of vaccine formulated from VT (A/Vietnam/1994/2004) strain, 1 at Day 0 and 1 at Day 21 and a 3rd dose of vaccine including VT strain at Month 6. The vaccine was administered in the deltoid region of the non-dominant arm.
- GSK1562902A V/I/12 Group: Healthy male or female subjects, between and including 18 and 60 years of age, who received 1 dose of vaccine formulated from VT (A/Vietnam/1994/2004) strain at Day 0 and 1 dose of the vaccine including IN (A/Indonesia/05/2005) strain at Month 12. The vaccine was administered in the deltoid region of the non-dominant arm.
- GSK1562902A V/V/12 Group: Healthy male or female subjects, between and including 18 and 60 years of age, who received 2 doses of vaccine formulated from VT (A/Vietnam/1994/2004) strain, 1 at Day 0 and 1 at Month 12. The vaccine was administered in the deltoid region of the non-dominant arm.
- GSK1562902A 2V/I/12 Group: Healthy male or female subjects, between and including 18 and 60 years of age, who received 2 doses of vaccine formulated from VT (A/Vietnam/1994/2004) strain, 1 at Day 0 and 1 at Day 21 and a 3rd dose of vaccine including IN (A/Indonesia/05/2005) strain at Month 12.The vaccine was administered in the deltoid region of the non-dominant arm.
- GSK1562902A 2V/V/12 Group: Healthy male or female subjects, between and including 18 and 60 years of age, who received 2 doses of vaccine formulated from VT (A/Vietnam/1994/2004) strain, 1 at Day 0 and 1 at Day 21 and a 3rd dose of vaccine including VT strain at Month 12.The vaccine was administered in the deltoid region of the non-dominant arm.
Period: Overall Study
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group | GSK1562902A V/I/12 Group | GSK1562902A V/V/12 Group | GSK1562902A 2V/I/12 Group | GSK1562902A 2V/V/12 Group
Started | 63 | 66 | 64 | 63 | 64 | 64 | 65 | 63
Completed | 52 | 57 | 61 | 55 | 59 | 59 | 55 | 51
Not Completed | 11 | 9 | 3 | 8 | 5 | 5 | 10 | 12
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Not completed — Lost to Follow-up | 7 | 8 | 3 | 5 | 5 | 2 | 8 | 10
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Vaccine Expired | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 3 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- GSK1562902A 2V/V/12 Group: Healthy male or female subjects, between and including 18 and 60 years of age, who received 2 doses of vaccine formulated from VT (A/Vietnam/1994/2004) strain, 1 at Day 0 and 1 at Day 21 and a 3rd dose of vaccine including VT strain at Month 12. The vaccine was administered in the deltoid region of the non-dominant arm.
- Total: Total of all reporting groups
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group | GSK1562902A V/I/12 Group | GSK1562902A V/V/12 Group | GSK1562902A 2V/I/12 Group | GSK1562902A 2V/V/12 Group | Total
Number analyzed (Participants) | 63 | 66 | 64 | 63 | 64 | 64 | 65 | 63 | 512
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.6 (12.9) | 33.1 (11.4) | 33.8 (11.8) | 33.4 (12.4) | 34.6 (12.9) | 34.8 (12.9) | 33.2 (11.2) | 34.3 (11.6) | 34.0 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 35 | 33 | 37 | 37 | 27 | 36 | 36 | 273
  Male | 31 | 31 | 31 | 26 | 27 | 37 | 29 | 27 | 239
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian / European heritage | 63 | 64 | 62 | 61 | 64 | 61 | 63 | 62 | 500
  Others | 0 | 2 | 2 | 2 | 0 | 3 | 2 | 1 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With H5N1 Haemagglutination-inhibition (HI) Antibody Concentrations Above the Cut-off Value
Description: The seropositivity cut-off for the assay was an antibody titer equal to or above (≥) 1:10, in the sera of subjects seronegative before vaccination. The flu strains assessed were A/Indonesia/05/2005 and A/Vietnam/1194/2004, for adults who received the booster dose at Month 6.
Time Frame: At Day 0
Population: This analysis was performed on the According-to-Protocol (ATP) Cohort for Immunogenicity, which included all evaluable subjects for whom immunogenicity data were available and who complied with the inclusion/exclusion criteria as defined in the protocol.
Measure: Count of Participants; unit: Participants
Groups:
- GSK1562902A 2V/I/6 Group: Healthy male or female subjects, between and including 18 and 60 years of age, who received 2 doses of vaccine formulated from VT (A/Vietnam/1994/2004) strain, 1 at Day 0 and 1 at Day 21 and a 3rd dose of vaccine including IN (A/Indonesia/05/2005) strain at Month 6. The vaccine was administered in the deltoid region of the non-dominant arm.
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 56 | 55 | 50 | 48
Participants
  A/Indonesia, Day 0 | 0 | 0 | 0 | 0
  A/Vietnam, Day 0 | 0 | 2 | 1 | 2

2. Primary Outcome: Number of Subjects With H5N1 Haemagglutination-inhibition (HI) Antibody Concentrations Above the Cut-off Value
Description: as for outcome 1
Time Frame: At Month 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 55 | 49 | 49 | 48
Participants
  A/Indonesia, Month 6 | 4 | 2 | 18 | 13
  A/Vietnam, Month 6 | 25 | 18 | 35 | 34

3. Primary Outcome: Number of Subjects With H5N1 Haemagglutination-inhibition (HI) Antibody Concentrations Above the Cut-off Value
Description: as for outcome 1
Time Frame: At Month 6 + 7 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 53 | 47 | 47 | 45
Participants
  A/Indonesia, Month 6 + 7 Days | 52 | 37 | 41 | 37
  A/Vietnam, Month 6 + 7 Days | 52 | 42 | 43 | 41

4. Primary Outcome: Number of Subjects With H5N1 Haemagglutination-inhibition (HI) Antibody Concentrations Above the Cut-off Value
Description: as for outcome 1
Time Frame: At Month 6 + 21 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 52 | 48 | 49 | 46
Participants
  A/Indonesia, Month 6 + 21 Days | 51 | 41 | 47 | 41
  A/Vietnam, Month 6 + 21 Days | 51 | 43 | 47 | 43

5. Primary Outcome: Geometric Mean Titers (GMTs) of H5N1 HI Antibodies
Description: GMTs were calculated for H5N1 HI antibodies against the A/Vietnam/1194/2004 or A/Indonesia/05/2005 strains, for the groups who received the booster dose at Month 6.
Time Frame: At Day 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 56 | 55 | 50 | 48
Titers
  A/Indonesia, Day 0 | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  A/Vietnam, Day 0 | 5.0 [5.0 to 5.0] | 5.3 [4.9 to 5.7] | 5.2 [4.8 to 5.7] | 5.7 [4.7 to 7.0]

6. Primary Outcome: Geometric Mean Titers (GMTs) of H5N1 HI Antibodies
Description: as for outcome 5
Time Frame: At Month 6
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 55 | 49 | 49 | 48
Titers
  A/Indonesia, Month 6 | 5.5 [5.0 to 6.0] | 5.3 [4.9 to 5.7] | 8.6 [6.6 to 11.3] | 7.2 [6.0 to 8.6]
  A/Vietnam, Month 6 | 12.0 [8.9 to 16.1] | 9.7 [7.4 to 12.7] | 29.9 [20.1 to 44.4] | 32.0 [21.3 to 48.0]

7. Primary Outcome: Geometric Mean Titers (GMTs) of H5N1 HI Antibodies
Description: as for outcome 5
Time Frame: At Month 6 + 7 Days
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 53 | 47 | 47 | 45
Titers
  A/Indonesia, Month 6 + 7 days | 152.9 [112.2 to 208.2] | 64.6 [41.3 to 101.1] | 120.0 [76.8 to 187.6] | 65.0 [42.1 to 100.2]
  A/Vietnam, Month 6 + 7 days | 226.3 [168.3 to 304.3] | 202.6 [130.7 to 314.1] | 182.7 [118.5 to 281.7] | 224.5 [144.9 to 347.7]

8. Primary Outcome: Geometric Mean Titers (GMTs) of H5N1 HI Antibodies
Description: as for outcome 5
Time Frame: At Month 6 + 21 Days
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 52 | 48 | 49 | 46
Titers
  A/Indonesia, Month 6 + 21 Days | 303.4 [215.7 to 426.6] | 92.4 [61.1 to 139.9] | 392.9 [256.7 to 601.4] | 127.7 [83.8 to 194.6]
  A/Vietnam, Month 6 + 21 Days | 434.7 [314.8 to 600.5] | 287.2 [180.3 to 457.5] | 571.4 [366.3 to 891.3] | 380.5 [240.2 to 602.9]

9. Primary Outcome: Seroconversion Factor for H5N1 Haemagglutination-inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: The seroconversion factor (SCF) was defined as the fold change in serum H5N1 HI geometric mean titers (GMTs) post-vaccination compared to Day 0. The 2 flu strains assessed were A/Vietnam/1194/2004 and A/Indonesia/5/2005, for adults who received the booster dose at Month 6.
Time Frame: At Month 6
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Increase
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 55 | 49 | 49 | 48
Fold Increase
  A/Indonesia, Month 6 | 1.1 [1.0 to 1.2] | 1.1 [1.0 to 1.1] | 1.7 [1.3 to 2.3] | 1.4 [1.2 to 1.7]
  A/Vietnam, Month 6 | 2.4 [1.8 to 3.2] | 1.8 [1.4 to 2.4] | 6.0 [4.0 to 8.9] | 5.6 [3.8 to 8.2]

10. Primary Outcome: Seroconversion Factor for H5N1 Haemagglutination-inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: as for outcome 9
Time Frame: At Month 6 + 7 Days
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Increase
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 53 | 47 | 47 | 45
Fold Increase
  A/Indonesia, Month 6 + 7 Days | 30.6 [22.4 to 41.6] | 12.9 [8.3 to 20.2] | 24.0 [15.4 to 37.5] | 13.0 [8.4 to 20.0]
  A/Vietnam, Month 6 + 7 Days | 45.3 [33.7 to 60.9] | 38.2 [23.7 to 56.3] | 36.5 [23.7 to 56.3] | 38.8 [24.7 to 60.9]

11. Primary Outcome: Seroconversion Factor for H5N1 Haemagglutination-inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: The seroconversion factor (SCF) was defined as the fold change in serum H5N1 HI geometric mean titers (GMTs) post vaccination compared to Day 0. The 2 flu strains assessed were A/Vietnam/1194/2004 and A/Indonesia/5/2005, for adults who received the booster dose at Month 6.
Time Frame: At Month 6 + 21 Days
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Increase
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 52 | 48 | 49 | 46
Fold Increase
  A/Indonesia, Month 6 + 21 Days | 60.7 [43.1 to 85.3] | 18.5 [12.2 to 28.0] | 78.6 [51.3 to 120.3] | 25.5 [16.8 to 38.9]
  A/Vietnam, Month 6 + 21 Days | 86.9 [63.0 to 120.1] | 54.2 [33.8 to 87.1] | 114.3 [73.3 to 178.3] | 66.0 [41.2 to 105.7]

12. Primary Outcome: Number of Seroconverted Subjects for H5N1 Haemagglutination-inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: A seroconverted (SCR) subject was defined as a vaccinated subject who had either a pre-vaccination titer < 1:10 and a post-vaccination titer ≥ 1:40 or a pre-vaccination titer ≥ 1:10 and at least a four-fold increase in post-vaccination titer. The 2 flu strains assessed were A/Vietnam/1194/2004 and A/Indonesia/5/2005, for adults who received the booster dose at Month 6.
Time Frame: At Month 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 55 | 49 | 49 | 48
Participants
  A/Indonesia, Month 6 | 0 | 0 | 5 | 2
  A/Vietnam, Month 6 | 14 | 6 | 26 | 27

13. Primary Outcome: Number of Seroconverted Subjects for H5N1 Haemagglutination-inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: as for outcome 12
Time Frame: At Month 6 + 7 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 53 | 47 | 47 | 45
Participants
  A/Indonesia, Month 6 + 7 Days | 49 | 35 | 40 | 33
  A/Vietnam, Month 6 + 7 Days | 52 | 42 | 42 | 39

14. Primary Outcome: Number of Seroconverted Subjects for H5N1 Haemagglutination-inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: as for outcome 12
Time Frame: At Month 6 + 21 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 52 | 48 | 49 | 46
Participants
  A/Indonesia, Month 6 + 21 Days | 51 | 40 | 46 | 40
  A/Vietnam, Month 6 + 21 Days | 51 | 43 | 46 | 42

15. Primary Outcome: Number of Seroprotected Subjects for H5N1 Haemagglutination-inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: A seroprotected (SPR) subject was defined as a vaccinated subject with serum H5N1 HI titer ≥ 1:40. The 2 flu strains assessed were A/Vietnam/1194/2004 and A/Indonesia/5/2005, for adults who received the booster dose at Month 6.
Time Frame: At Day 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 56 | 55 | 50 | 48
Participants
  A/Indonesia, Day 0 | 0 | 0 | 0 | 0
  A/Vietnam, Day 0 | 0 | 0 | 1 | 2

16. Primary Outcome: Number of Seroprotected Subjects for H5N1 Haemagglutination-inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: as for outcome 15
Time Frame: At Month 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 55 | 49 | 49 | 48
Participants
  A/Indonesia, Month 6 | 0 | 0 | 5 | 2
  A/Vietnam, Month 6 | 14 | 7 | 26 | 28

17. Primary Outcome: Number of Seroprotected Subjects for H5N1 Haemagglutination-inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: as for outcome 15
Time Frame: At Month 6 + 7 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 53 | 47 | 47 | 45
Participants
  A/Indonesia, Month 6 + 7 Days | 49 | 35 | 40 | 33
  A/Vietnam, Month 6 + 7 Days | 52 | 42 | 42 | 40

18. Primary Outcome: Number of Seroprotected Subjects for H5N1 Haemagglutination-inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: as for outcome 15
Time Frame: At Month 6 + 21 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 52 | 48 | 49 | 46
Participants
  A/Indonesia, Month 6 + 21 Days | 51 | 40 | 46 | 40
  A/Vietnam, Month 6 + 21 Days | 51 | 43 | 46 | 42

19. Primary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were ecchymosis, induration, pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 ecchymosis/induration/redness/swelling = spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses, up to 6/12 months + 7 days
Population: This analysis was performed on the Total vaccinated Cohort, which included all vaccinated subjects for whom data were available and who had their symptom sheets filled in. The data for Dose 3 were not collected from subjects who did not receive the booster dose, given at either Month 6 or Month 12.
Measure: Count of Participants; unit: Participants
Groups:
- GSK1562902A 2V/I/12 Group: Healthy male or female subjects, between and including 18 and 60 years of age, who received 2 doses of vaccine formulated from VT (A/Vietnam/1994/2004) strain, 1 at Day 0 and 1 at Day 21 and a 3rd dose of vaccine including IN (A/Indonesia/05/2005) strain at Month 12. The vaccine was administered in the deltoid region of the non-dominant arm.
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group | GSK1562902A V/I/12 Group | GSK1562902A V/V/12 Group | GSK1562902A 2V/I/12 Group | GSK1562902A 2V/V/12 Group
Number analyzed (Participants) | 62 | 66 | 64 | 62 | 64 | 64 | 65 | 63
Participants
  Any Ecchymosis, Dose 1 | 1 | 1 | 2 | 0 | 0 | 0 | 3 | 1
  Grade 3 Ecchymosis, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Induration, Dose 1 | 9 | 9 | 10 | 20 | 7 | 9 | 14 | 8
  Grade 3 Induration, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain, Dose 1 | 50 | 61 | 54 | 56 | 53 | 52 | 57 | 54
  Grade 3 Pain, Dose 1 | 2 | 2 | 0 | 4 | 5 | 5 | 2 | 1
  Any Redness, Dose 1 | 4 | 6 | 5 | 8 | 5 | 8 | 6 | 5
  Grade 3 Redness, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling, Dose 1 | 7 | 7 | 7 | 14 | 5 | 10 | 8 | 9
  Grade 3 Swelling, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Ecchymosis, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Any Ecchymosis, Dose 2 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 0
  Grade 3 Ecchymosis, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Grade 3 Ecchymosis, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Induration, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Any Induration, Dose 2 | 13 | 11 | 9 | 14 | 11 | 11 | 9 | 8
  Grade 3 Induration, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Grade 3 Induration, Dose 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Any Pain, Dose 2 | 46 | 49 | 50 | 49 | 54 | 47 | 49 | 47
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Grade 3 Pain, Dose 2 | 4 | 4 | 0 | 4 | 4 | 3 | 0 | 1
  Any Redness, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Any Redness, Dose 2 | 9 | 8 | 11 | 7 | 5 | 7 | 7 | 8
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Grade 3 Redness, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Any Swelling, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Any Swelling, Dose 2 | 7 | 12 | 10 | 10 | 6 | 7 | 4 | 10
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Grade 3 Swelling, Dose 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Ecchymosis, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Any Ecchymosis, Dose 3 |  |  | 0 | 0 |  |  | 0 | 0
  Grade 3 Ecchymosis, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Grade 3 Ecchymosis, Dose 3 |  |  | 0 | 0 |  |  | 0 | 0
  Any Induration, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Any Induration, Dose 3 |  |  | 16 | 13 |  |  | 15 | 10
  Grade 3 Induration, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Grade 3 Induration, Dose 3 |  |  | 0 | 0 |  |  | 0 | 0
  Any Pain, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Any Pain, Dose 3 |  |  | 53 | 51 |  |  | 48 | 44
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Grade 3 Pain, Dose 3 |  |  | 5 | 5 |  |  | 4 | 4
  Any Redness, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Any Redness, Dose 3 |  |  | 8 | 7 |  |  | 8 | 8
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Grade 3 Redness, Dose 3 |  |  | 0 | 0 |  |  | 0 | 0
  Any Swelling, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Any Swelling, Dose 3 |  |  | 15 | 13 |  |  | 10 | 8
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Grade 3 Swelling, Dose 3 |  |  | 0 | 0 |  |  | 0 | 0
  Any Ecchymosis, Across doses | 2 | 1 | 2 | 1 | 0 | 2 | 4 | 1
  Grade 3 Ecchymosis, Across doses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Induration, Across doses | 17 | 13 | 22 | 25 | 14 | 16 | 24 | 19
  Grade 3 Induration, Across doses | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain, Across doses | 56 | 62 | 61 | 59 | 61 | 57 | 62 | 58
  Grade 3 Pain, Across doses | 6 | 6 | 5 | 10 | 8 | 8 | 5 | 5
  Any Redness, Across doses | 11 | 8 | 16 | 13 | 8 | 11 | 13 | 15
  Grade 3 Redness, Across doses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Any Swelling, Across doses | 12 | 15 | 21 | 22 | 10 | 13 | 16 | 16
  Grade 3 Swelling, Across doses | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

20. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, fever [defined as axillary temperature above (>) 38 degrees Celsius (°C)], headache, myalgia, shivering and sweating. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 40.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses, up to 12 months + 7 days
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group | GSK1562902A V/I/12 Group | GSK1562902A V/V/12 Group | GSK1562902A 2V/I/12 Group | GSK1562902A 2V/V/12 Group
Number analyzed (Participants) | 62 | 66 | 64 | 62 | 64 | 64 | 65 | 63
Participants
  Any Arthralgia, Dose 1 | 8 | 12 | 11 | 15 | 13 | 9 | 8 | 6
  Grade 3 Arthralgia, Dose 1 | 2 | 1 | 0 | 0 | 2 | 0 | 1 | 0
  Related Arthralgia, Dose 1 | 7 | 12 | 9 | 12 | 13 | 8 | 6 | 6
  Any Fatigue, Dose 1 | 25 | 27 | 24 | 26 | 27 | 21 | 25 | 25
  Grade 3 Fatigue, Dose 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0
  Related Fatigue, Dose 1 | 24 | 25 | 20 | 20 | 27 | 19 | 19 | 23
  Any Fever, Dose 1 | 4 | 3 | 0 | 1 | 0 | 1 | 1 | 2
  Grade 3 Fever, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Fever, Dose 1 | 4 | 3 | 0 | 0 | 0 | 0 | 1 | 2
  Any Headache, Dose 1 | 22 | 18 | 19 | 25 | 18 | 24 | 28 | 20
  Grade 3 Headache, Dose 1 | 3 | 0 | 0 | 4 | 0 | 1 | 0 | 1
  Related Headache, Dose 1 | 21 | 15 | 18 | 21 | 17 | 21 | 23 | 19
  Any Myalgia, Dose 1 | 29 | 29 | 31 | 32 | 31 | 29 | 27 | 31
  Grade 3 Myalgia, Dose 1 | 3 | 1 | 0 | 0 | 2 | 1 | 2 | 0
  Related Myalgia, Dose 1 | 29 | 26 | 29 | 30 | 30 | 27 | 26 | 29
  Any Shivering, Dose 1 | 13 | 12 | 10 | 21 | 15 | 8 | 9 | 14
  Grade 3 Shivering, Dose 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Related Shivering, Dose 1 | 13 | 11 | 8 | 19 | 14 | 8 | 6 | 13
  Any Sweating, Dose 1 | 6 | 7 | 9 | 12 | 5 | 2 | 5 | 12
  Grade 3 Sweating, Dose 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Related Sweating, Dose 1 | 5 | 7 | 8 | 10 | 5 | 1 | 4 | 12
  Any Arthralgia, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Any Arthralgia, Dose 2 | 12 | 20 | 11 | 13 | 14 | 12 | 15 | 15
  Grade 3 Arthralgia, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Grade 3 Arthralgia, Dose 2 | 1 | 1 | 0 | 1 | 1 | 1 | 3 | 1
  Related Arthralgia, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Related Arthralgia, Dose 2 | 12 | 16 | 9 | 12 | 14 | 11 | 13 | 14
  Any Fatigue, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Any Fatigue, Dose 2 | 23 | 27 | 28 | 21 | 30 | 22 | 21 | 27
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Grade 3 Fatigue, Dose 2 | 2 | 1 | 0 | 0 | 5 | 3 | 4 | 0
  Related Fatigue, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Related Fatigue, Dose 2 | 20 | 24 | 25 | 19 | 28 | 22 | 18 | 26
  Any Fever, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Any Fever, Dose 2 | 2 | 2 | 1 | 0 | 4 | 3 | 1 | 2
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Grade 3 Fever, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Fever, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Related Fever, Dose 2 | 2 | 2 | 1 | 0 | 4 | 2 | 1 | 2
  Any Headache, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Any Headache, Dose 2 | 22 | 22 | 24 | 26 | 24 | 22 | 20 | 15
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Grade 3 Headache, Dose 2 | 1 | 2 | 0 | 3 | 1 | 2 | 1 | 0
  Related Headache, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Related Headache, Dose 2 | 18 | 19 | 18 | 22 | 23 | 20 | 16 | 13
  Any Myalgia, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Any Myalgia, Dose 2 | 28 | 32 | 27 | 22 | 40 | 30 | 29 | 28
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Grade 3 Myalgia, Dose 2 | 2 | 2 | 0 | 1 | 3 | 2 | 3 | 2
  Related Myalgia, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Related Myalgia, Dose 2 | 25 | 27 | 23 | 21 | 37 | 26 | 28 | 25
  Any Shivering, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Any Shivering, Dose 2 | 14 | 21 | 10 | 13 | 17 | 14 | 9 | 14
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Grade 3 Shivering, Dose 2 | 3 | 2 | 1 | 1 | 4 | 2 | 2 | 0
  Related Shivering, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Related Shivering, Dose 2 | 12 | 19 | 9 | 13 | 17 | 14 | 8 | 14
  Any Sweating, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Any Sweating, Dose 2 | 10 | 12 | 12 | 5 | 13 | 6 | 12 | 7
  Grade 3 Sweating, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Grade 3 Sweating, Dose 2 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 0
  Related Sweating, Dose 2: number analyzed (Participants) | 57 | 57 | 64 | 61 | 62 | 58 | 63 | 60
  Related Sweating, Dose 2 | 8 | 9 | 12 | 4 | 12 | 6 | 10 | 6
  Any Arthralgia, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Any Arthralgia, Dose 3 |  |  | 18 | 19 |  |  | 19 | 14
  Grade 3 Arthralgia, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Grade 3 Arthralgia, Dose 3 |  |  | 0 | 3 |  |  | 4 | 1
  Related Arthralgia, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Related Arthralgia, Dose 3 |  |  | 17 | 16 |  |  | 17 | 13
  Any Fatigue, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Any Fatigue, Dose 3 |  |  | 32 | 30 |  |  | 29 | 29
  Grade 3 Fatigue, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Grade 3 Fatigue, Dose 3 |  |  | 2 | 3 |  |  | 0 | 2
  Related Fatigue, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Related Fatigue, Dose 3 |  |  | 28 | 27 |  |  | 24 | 28
  Any Fever, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Any Fever, Dose 3 |  |  | 3 | 3 |  |  | 3 | 2
  Grade 3 Fever, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Grade 3 Fever, Dose 3 |  |  | 0 | 0 |  |  | 0 | 0
  Related Fever, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Related Fever, Dose 3 |  |  | 2 | 3 |  |  | 3 | 2
  Any Headache, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Any Headache, Dose 3 |  |  | 30 | 28 |  |  | 23 | 32
  Grade 3 Headache, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Grade 3 Headache, Dose 3 |  |  | 1 | 4 |  |  | 1 | 2
  Related Headache, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Related Headache, Dose 3 |  |  | 22 | 26 |  |  | 20 | 25
  Any Myalgia, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Any Myalgia, Dose 3 |  |  | 35 | 36 |  |  | 31 | 29
  Grade 3 Myalgia, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Grade 3 Myalgia, Dose 3 |  |  | 2 | 3 |  |  | 4 | 2
  Related Myalgia, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Related Myalgia, Dose 3 |  |  | 31 | 33 |  |  | 28 | 27
  Any Shivering, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Any Shivering, Dose 3 |  |  | 17 | 19 |  |  | 18 | 21
  Grade 3 Shivering, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Grade 3 Shivering, Dose 3 |  |  | 3 | 4 |  |  | 2 | 3
  Related Shivering, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Related Shivering, Dose 3 |  |  | 15 | 17 |  |  | 17 | 21
  Any Sweating, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Any Sweating, Dose 3 |  |  | 13 | 13 |  |  | 11 | 15
  Grade 3 Sweating, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Grade 3 Sweating, Dose 3 |  |  | 1 | 2 |  |  | 1 | 0
  Related Sweating, Dose 3: number analyzed (Participants) | 0 | 0 | 63 | 58 | 0 | 0 | 55 | 52
  Related Sweating, Dose 3 |  |  | 11 | 12 |  |  | 10 | 13
  Any Arthralgia, Across doses | 17 | 25 | 27 | 28 | 20 | 13 | 29 | 26
  Grade 3 Arthralgia, Across doses | 3 | 2 | 0 | 4 | 3 | 1 | 5 | 2
  Related Arthralgia, Across doses | 16 | 22 | 26 | 25 | 20 | 12 | 25 | 24
  Any Fatigue, Across doses | 35 | 37 | 45 | 44 | 37 | 33 | 47 | 44
  Grade 3 Fatigue, Across doses | 2 | 2 | 3 | 3 | 5 | 4 | 4 | 2
  Related Fatigue, Across doses | 33 | 34 | 42 | 38 | 36 | 31 | 40 | 42
  Any Fever, Across doses | 6 | 4 | 4 | 4 | 4 | 4 | 4 | 5
  Grade 3 Fever, Across doses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Fever, Across doses | 6 | 4 | 3 | 3 | 4 | 2 | 4 | 5
  Any Headache, Across doses | 34 | 31 | 41 | 41 | 31 | 34 | 45 | 41
  Grade 3 Headache, Across doses | 4 | 2 | 1 | 8 | 1 | 3 | 2 | 3
  Related Headache, Across doses | 31 | 28 | 36 | 38 | 30 | 30 | 41 | 35
  Any Myalgia, Across doses | 41 | 41 | 47 | 48 | 49 | 41 | 45 | 47
  Grade 3 Myalgia, Across doses | 5 | 3 | 2 | 4 | 4 | 3 | 7 | 4
  Related Myalgia, Across doses | 39 | 38 | 46 | 47 | 45 | 39 | 43 | 43
  Any Shivering, Across doses | 22 | 28 | 24 | 36 | 22 | 19 | 25 | 29
  Grade 3 Shivering, Across doses | 6 | 3 | 3 | 5 | 4 | 2 | 4 | 4
  Related Shivering, Across doses | 21 | 26 | 21 | 34 | 22 | 19 | 23 | 29
  Any Sweating, Across doses | 15 | 18 | 23 | 20 | 16 | 7 | 23 | 25
  Grade 3 Sweating, Across doses | 1 | 1 | 1 | 3 | 1 | 1 | 3 | 1
  Related Sweating, Across doses | 13 | 15 | 21 | 17 | 15 | 6 | 21 | 24

21. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 30-day (Days 0-29) post-primary vaccination period (Month 6 + 30 days)
Population: This analysis was performed on the Total vaccinated Cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group | GSK1562902A V/I/12 Group | GSK1562902A V/V/12 Group | GSK1562902A 2V/I/12 Group | GSK1562902A 2V/V/12 Group
Number analyzed (Participants) | 63 | 66 | 64 | 63 | 64 | 64 | 65 | 63
Participants
  Any AEs | 31 | 19 | 32 | 28 | 18 | 10 | 19 | 24
  Grade 3 AEs | 3 | 4 | 2 | 3 | 0 | 2 | 1 | 7
  Related AEs | 12 | 11 | 11 | 15 | 5 | 3 | 6 | 6

22. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: as for outcome 21
Time Frame: During the 30-day (Days 0-29) post-booster vaccination period (Month 12 + 30 days)
Population: This analysis was performed on the Total vaccinated Cohort, which included all vaccinated subjects for whom data were available. Data were collected only for subjects who received the Month 12 vaccine dose.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group | GSK1562902A V/I/12 Group | GSK1562902A V/V/12 Group | GSK1562902A 2V/I/12 Group | GSK1562902A 2V/V/12 Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 62 | 58 | 56 | 53
Participants
  Any AE(s) |  |  |  |  | 16 | 10 | 16 | 14
  Grade 3 AE(s) |  |  |  |  | 2 | 2 | 2 | 1
  Related AE(s) |  |  |  |  | 7 | 4 | 9 | 9

23. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: as for outcome 21
Time Frame: During the entire study period (Day 0 to Month 18)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group | GSK1562902A V/I/12 Group | GSK1562902A V/V/12 Group | GSK1562902A 2V/I/12 Group | GSK1562902A 2V/V/12 Group
Number analyzed (Participants) | 63 | 66 | 64 | 63 | 64 | 64 | 65 | 63
Participants | 35 | 23 | 32 | 31 | 27 | 24 | 30 | 31

24. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (Day 0 to Month 18)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group | GSK1562902A V/I/12 Group | GSK1562902A V/V/12 Group | GSK1562902A 2V/I/12 Group | GSK1562902A 2V/V/12 Group
Number analyzed (Participants) | 63 | 66 | 64 | 63 | 64 | 64 | 65 | 63
Participants | 4 | 1 | 0 | 3 | 1 | 5 | 1 | 3

25. Primary Outcome: Number of Booster Seroconverted Subjects Against 2 Strains of Influenza Disease
Description: Booster seroconversion (SCR) was defined as: For seronegative subjects at pre-booster (Month 6), antibody titer ≥ 1:40 at Month 6 + 7 days; For seropositive subjects at pre-booster (Month 6), antibody titer at Month 6 + 7 days ≥ 4 fold the pre-vaccination antibody titer at Month 6. The 2 flu strains assessed were A/Vietnam/1194/2004 and A/Indonesia/5/2005, for adults who received the booster dose at Month 6.
Time Frame: At Month 6 + 7 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 53 | 47 | 47 | 45
Participants
  A/Indonesia, Month 6 + 7 Days | 48 | 35 | 40 | 31
  A/Vietnam, Month 6 + 7 Days | 47 | 40 | 31 | 30

26. Primary Outcome: Number of Booster Seroconverted Subjects Against 2 Strains of Influenza Disease
Description: Booster SCR was defined as: For seronegative subjects at pre-booster (Month 6), antibody titer ≥ 1:40 at Month 6 + 7 days; For seropositive subjects at pre-booster (Month 6), antibody titer at Month 6 + 7 days ≥ 4 fold the pre-vaccination antibody titer at Month 6. The 2 flu strains assessed were A/Vietnam/1194/2004 and A/Indonesia/5/2005, for adults who received the booster dose at Month 6.
Time Frame: At Month 6 + 21 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 52 | 48 | 49 | 46
Participants
  A/Indonesia, Month 6 + 21 Days | 51 | 39 | 45 | 39
  A/Vietnam, Month 6 + 21 Days | 51 | 42 | 44 | 38

27. Primary Outcome: Booster Factor of H5N1 HI Antibodies Against 2 Strains of Influenza Disease
Description: Booster Factor (Seroconversion Factor booster) was defined as the fold change in H5N1 HI antibodies between the pre- and post-booster vaccination time-points (mean[log10(POST/M6)]). The 2 flu strains assessed were A/Vietnam/1194/2004 and A/Indonesia/05/2005, for groups who received the booster dose at Month 6.
Time Frame: At Month 6 + 7 Days
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Increase
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 53 | 47 | 47 | 45
Fold Increase
  A/Indonesia, Month 6 + 7 Days | 27.9 [20.4 to 38.3] | 12.3 [7.8 to 19.2] | 14.5 [8.7 to 24.3] | 9.2 [6.2 to 13.7]
  A/Vietnam, Month 6 + 7 Days | 18.2 [12.8 to 26.0] | 20.3 [12.7 to 32.5] | 6.3 [4.1 to 9.7] | 6.9 [4.5 to 10.7]

28. Primary Outcome: Booster Factor of H5N1 HI Antibodies Against 2 Strains of Influenza Disease
Description: as for outcome 27
Time Frame: At Month 6 + 21 Days
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Increase
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 52 | 48 | 49 | 46
Fold Increase
  A/Indonesia, Month 6 + 21 Days | 55.3 [39.5 to 77.4] | 17.6 [11.5 to 26.8] | 45.6 [30.8 to 67.4] | 17.9 [11.9 to 27.0]
  A/Vietnam, Month 6 + 21 Days | 35.4 [24.5 to 51.1] | 29.2 [18.2 to 46.6] | 19.1 [12.4 to 29.4] | 11.5 [7.3 to 18.0]

29. Secondary Outcome: GMTs of H5N1 HI Antibodies Against 2 Strains of Influenza Disease for Groups Who Received Booster Dose at Month 12
Description: GMTs were calculated for H5N1 HI antibodies against the A/Vietnam/1194/2004 or A/Indonesia/05/2005 strains.
Time Frame: At Day 0, Day 21, Day 42, Month 6, Month 12, Month 12 + 7 Days, Month 12 + 21 Days and at Month 18
Population: This analysis was performed on the ATP Cohort for Immunogenicity and ATP Cohort for Persistence (only for Month 18), which included all evaluable subjects for whom immunogenicity were available and who complied with the inclusion/exclusion criteria defined in the protocol. Day 42 data were available only from subjects who received 3 vaccine doses.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK1562902A V/I/12 Group | GSK1562902A V/V/12 Group | GSK1562902A 2V/I/12 Group | GSK1562902A 2V/V/12 Group
Number analyzed (Participants) | 59 | 60 | 55 | 55
Titers
  A/Indonesia, Day 0 | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  A/Indonesia, Day 21: number analyzed (Participants) | 58 | 60 | 55 | 55
  A/Indonesia, Day 21 | 6.8 [5.5 to 8.3] | 6.3 [5.2 to 7.7] | 6.0 [5.2 to 6.8] | 5.3 [5.0 to 5.7]
  A/Indonesia, Day 42: number analyzed (Participants) | 0 | 0 | 49 | 48
  A/Indonesia, Day 42 |  |  | 28.0 [18.0 to 43.6] | 18.6 [12.7 to 27.2]
  A/Indonesia, Month 6: number analyzed (Participants) | 59 | 57 | 52 | 51
  A/Indonesia, Month 6 | 5.7 [5.1 to 6.4] | 5.4 [4.8 to 6.0] | 10.2 [7.8 to 13.3] | 6.5 [5.6 to 7.5]
  A/Indonesia, Month 12: number analyzed (Participants) | 52 | 52 | 41 | 44
  A/Indonesia, Month 12 | 5.8 [5.0 to 6.8] | 5.9 [5.1 to 6.8] | 5.7 [5.0 to 6.5] | 8.4 [6.4 to 11.1]
  A/Indonesia, Month 12 + 7 Days: number analyzed (Participants) | 50 | 51 | 40 | 43
  A/Indonesia, Month 12 + 7 Days | 97.8 [66.5 to 143.8] | 196.2 [128.6 to 299.2] | 106.5 [66.7 to 170.0] | 239.4 [149.9 to 382.2]
  A/Indonesia, Month 12 + 21 Days: number analyzed (Participants) | 50 | 51 | 40 | 43
  A/Indonesia, Month 12 + 21 Days | 139.3 [92.0 to 211.0] | 420.0 [283.8 to 621.6] | 191.9 [121.6 to 303.0] | 624.9 [469.3 to 831.9]
  A/Indonesia, Month 18: number analyzed (Participants) | 45 | 49 | 39 | 40
  A/Indonesia, Month 18 | 139.3 [85.7 to 226.6] | 56.6 [35.5 to 90.2] | 385.9 [252.9 to 588.6] | 121.3 [76.6 to 192.0]
  A/Vietnam, Day 0 | 5.0 [5.0 to 5.0] | 5.1 [4.9 to 5.4] | 5.1 [4.9 to 5.4] | 5.2 [4.8 to 5.5]
  A/Vietnam, Day 21: number analyzed (Participants) | 58 | 60 | 55 | 55
  A/Vietnam, Day 21 | 22.1 [14.5 to 33.8] | 17.6 [12.3 to 25.2] | 21.4 [14.3 to 32.0] | 15.8 [10.9 to 23.1]
  A/Vietnam, Day 42: number analyzed (Participants) | 0 | 0 | 49 | 48
  A/Vietnam, Day 42 |  |  | 239.4 [157.2 to 364.8] | 178.3 [116.6 to 272.5]
  A/Vietnam, Month 6: number analyzed (Participants) | 59 | 57 | 52 | 51
  A/Vietnam, Month 6 | 13.2 [9.3 to 18.7] | 10.6 [8.0 to 14.0] | 38.4 [26.6 to 55.5] | 24.0 [17.2 to 33.5]
  A/Vietnam, Month 12: number analyzed (Participants) | 52 | 52 | 41 | 44
  A/Vietnam, Month 12 | 8.4 [6.4 to 11.0] | 9.9 [7.3 to 13.5] | 14.2 [10.1 to 20.1] | 17.4 [11.6 to 25.9]
  A/Vietnam, Month 12 + 7 Days: number analyzed (Participants) | 50 | 51 | 40 | 43
  A/Vietnam, Month 12 + 7 Days | 235.9 [153.7 to 362.1] | 354.3 [244.7 to 513.0] | 257.7 [162.4 to 409.0] | 358.2 [228.7 to 561.1]
  A/Vietnam, Month 12 + 21 Days: number analyzed (Participants) | 50 | 51 | 40 | 43
  A/Vietnam, Month 12 + 21 Days | 352.6 [229.9 to 540.8] | 662.2 [458.3 to 956.6] | 441.0 [279.5 to 695.9] | 942.2 [703.1 to 1262.7]
  A/Vietnam, Month 18: number analyzed (Participants) | 45 | 49 | 39 | 40
  A/Vietnam, Month 18 | 115.8 [71.9 to 186.3] | 76.1 [47.1 to 123.1] | 337.5 [219.5 to 518.9] | 149.3 [93.0 to 239.6]

30. Secondary Outcome: Number of Seroconverted Subjects for H5N1 HI Antibodies Against 2 Strains of Influenza Disease, for Groups Who Received Booster Dose at Month 12
Description: A seroconverted (SCR) subject was defined as a vaccinated subject who had either a pre-vaccination titer < 1:10 and a post-vaccination titer ≥ 1:40 or a pre-vaccination titer ≥ 1:10 and at least a four-fold increase in post-vaccination titer. The 2 flu strains assessed were A/Vietnam/1194/2004 and A/Indonesia/5/2005.
Time Frame: At Day 21, Day 42, Month 6, Month 12, Month 12 + 7 Days, Month 12 + 21 Days
Population: This analysis was performed on the ATP Cohort for Immunogenicity, which included all evaluable subjects for whom immunogenicity data were available and who complied with the inclusion/exclusion criteria as defined in the protocol. Day 42 data were available only from subjects who received 3 vaccine doses.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/12 Group | GSK1562902A V/V/12 Group | GSK1562902A 2V/I/12 Group | GSK1562902A 2V/V/12 Group
Number analyzed (Participants) | 59 | 60 | 55 | 55
Participants
  A/Indonesia, Day 21: number analyzed (Participants) | 58 | 60 | 55 | 55
  A/Indonesia, Day 21 | 5 | 3 | 1 | 0
  A/Indonesia, Day 42: number analyzed (Participants) | 0 | 0 | 49 | 48
  A/Indonesia, Day 42 |  |  | 24 | 20
  A/Indonesia, Month 6: number analyzed (Participants) | 59 | 57 | 52 | 51
  A/Indonesia, Month 6 | 0 | 1 | 7 | 1
  A/Indonesia, Month 12: number analyzed (Participants) | 52 | 52 | 41 | 44
  A/Indonesia, Month 12 | 6 | 2 | 0 | 5
  A/Indonesia, Month 12 + 7 Days: number analyzed (Participants) | 50 | 51 | 40 | 43
  A/Indonesia, Month 12 + 7 Days | 40 | 44 | 34 | 39
  A/Indonesia, Month 12 + 21 Days: number analyzed (Participants) | 50 | 51 | 40 | 43
  A/Indonesia, Month 12 + 21 Days | 42 | 49 | 36 | 43
  A/Vietnam, Day 21: number analyzed (Participants) | 58 | 60 | 55 | 55
  A/Vietnam, Day 21 | 26 | 24 | 25 | 16
  A/Vietnam, Day 42: number analyzed (Participants) | 0 | 0 | 49 | 48
  A/Vietnam, Day 42 |  |  | 44 | 43
  A/Vietnam, Month 6: number analyzed (Participants) | 59 | 57 | 52 | 51
  A/Vietnam, Month 6 | 15 | 10 | 35 | 24
  A/Vietnam, Month 12: number analyzed (Participants) | 52 | 52 | 41 | 44
  A/Vietnam, Month 12 | 6 | 10 | 9 | 17
  A/Vietnam, Month 12 + 7 Days: number analyzed (Participants) | 50 | 51 | 40 | 43
  A/Vietnam, Month 12 + 7 Days | 45 | 49 | 37 | 40
  A/Vietnam, Month 12 + 21 Days: number analyzed (Participants) | 50 | 51 | 40 | 43
  A/Vietnam, Month 12 + 21 Days | 46 | 50 | 38 | 43

31. Secondary Outcome: Number of Seroconverted Subjects for H5N1 HI Antibodies Against 2 Strains of Influenza Disease, for Groups Who Received Booster Dose at Month 12
Description: Seroconversion defined as: For initially seronegative subjects, antibody titer ≥ 1:40 after vaccination; For initially seropositive subjects, antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer. The 2 flu strains assessed were A/Vietnam/1194/2004 and A/Indonesia/05/2005.
Time Frame: At Month 12 + 7 Days, Month 12 + 21 Days and Month 18
Population: This analysis was performed on the According-to-Protocol (ATP) Cohort for Persistence, which included all evaluable subjects for whom ilong term immunogenicity data were available and who complied with the inclusion/exclusion criteria as defined in the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/12 Group | GSK1562902A V/V/12 Group | GSK1562902A 2V/I/12 Group | GSK1562902A 2V/V/12 Group
Number analyzed (Participants) | 47 | 48 | 40 | 40
Participants
  A/Indonesia, Month 12 + 7 Days | 40 | 37 | 36 | 34
  A/Indonesia, Month 12 + 21 Days | 46 | 39 | 40 | 36
  A/Indonesia, Month 18: number analyzed (Participants) | 44 | 48 | 39 | 40
  A/Indonesia, Month 18 | 39 | 34 | 37 | 34
  A/Vietnam, Month 12 + 7 Days | 43 | 41 | 35 | 34
  A/Vietnam, Month 12 + 21 Days | 47 | 42 | 40 | 37
  A/Vietnam, Month 18: number analyzed (Participants) | 44 | 48 | 39 | 40
  A/Vietnam, Month 18 | 30 | 33 | 34 | 29

32. Secondary Outcome: Seroconversion Factor for H5N1 HI Antibodies Against 2 Strains of Influenza Disease, for Groups Who Received the Booster Dose at Month 12
Description: The seroconversion factor (SCF) was defined as the fold change in serum hemagglutination inhibition (HI) geometric mean titers (GMTs) post-vaccination compared to Day 0. The 2 flu strains assessed were A/Vietnam/1194/2004 and A/Indonesia/5/2005.
Time Frame: At Day 21, Day 42, Month 6, Month 12, Month 12 + 7 Days, Month 12 + 21 Days
Population: This analysis was performed on the According-to-Protocol (ATP) Cohort for Immunogenicity, which included all evaluable subjects for whom immunogenicity data were available and who complied with the inclusion/exclusion criteria as defined in the protocol. Day 42 data were available only from subjects who received 3 vaccine doses.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Increase
Arm/Group | GSK1562902A V/I/12 Group | GSK1562902A V/V/12 Group | GSK1562902A 2V/I/12 Group | GSK1562902A 2V/V/12 Group
Number analyzed (Participants) | 59 | 57 | 52 | 51
Fold Increase
  A/Indonesia, Day 21: number analyzed (Participants) | 53 | 55 | 48 | 49
  A/Indonesia, Day 21 | 1.4 [1.1 to 1.7] | 1.3 [1.0 to 1.6] | 1.2 [1.0 to 1.3] | 1.1 [1.0 to 1.2]
  A/Indonesia, Day 42: number analyzed (Participants) | 0 | 0 | 42 | 43
  A/Indonesia, Day 42 |  |  | 5.9 [3.6 to 9.5] | 3.6 [2.5 to 5.3]
  A/Indonesia, Month 6 | 1.1 [1.0 to 1.3] | 1.1 [1.0 to 1.2] | 2.0 [1.6 to 2.7] | 1.3 [1.1 to 1.5]
  A/Indonesia, Month 12: number analyzed (Participants) | 52 | 52 | 44 | 41
  A/Indonesia, Month 12 | 1.2 [1.0 to 1.2] | 1.2 [1.0 to 1.2] | 1.7 [1.3 to 2.2] | 1.1 [1.0 to 1.3]
  A/Indonesia, Month 12 + 7 Days: number analyzed (Participants) | 51 | 50 | 43 | 40
  A/Indonesia, Month 12 + 7 Days | 39.2 [25.7 to 59.8] | 19.6 [13.3 to 28.8] | 47.9 [30.0 to 76.4] | 21.3 [13.3 to 34.0]
  A/Indonesia, Month 12 + 21 Days: number analyzed (Participants) | 51 | 50 | 43 | 40
  A/Indonesia, Month 12 + 21 Days | 84.0 [56.8 to 124.3] | 27.9 [18.4 to 42.2] | 125.0 [93.9 to 166.4] | 38.4 [24.3 to 60.6]
  A/Vietnam, Day 21: number analyzed (Participants) | 53 | 55 | 48 | 49
  A/Vietnam, Day 21 | 4.1 [2.6 to 6.3] | 3.6 [2.5 to 5.2] | 3.8 [2.5 to 5.6] | 3.2 [2.2 to 4.8]
  A/Vietnam, Day 42: number analyzed (Participants) | 0 | 0 | 42 | 43
  A/Vietnam, Day 42 |  |  | 45.6 [28.4 to 73.4] | 34.4 [22.7 to 52.2]
  A/Vietnam, Month 6 | 2.6 [1.9 to 3.7] | 2.1 [1.6 to 2.7] | 7.5 [5.2 to 10.8] | 4.6 [3.4 to 6.4]
  A/Vietnam, Month 12: number analyzed (Participants) | 52 | 52 | 44 | 41
  A/Vietnam, Month 12 | 2.0 [1.5 to 2.7] | 1.6 [1.3 to 2.1] | 3.5 [2.3 to 5.2] | 2.7 [1.9 to 3.9]
  A/Vietnam, Month 12 + 7 Days: number analyzed (Participants) | 51 | 50 | 43 | 40
  A/Vietnam, Month 12 + 7 Days | 70.9 [48.9 to 102.6] | 45.9 [29.8 to 70.7] | 71.6 [45.7 to 112.2] | 49.4 [31.0 to 78.6]
  A/Vietnam, Month 12 + 21 Days: number analyzed (Participants) | 51 | 50 | 43 | 40
  A/Vietnam, Month 12 + 21 Days | 132.4 [91.7 to 191.3] | 68.6 [44.5 to 105.8] | 188.4 [140.6 to 252.5] | 84.5 [53.3 to 133.9]

33. Secondary Outcome: Number of Seroprotected Subjects for H5N1 HI Antibodies Against 2 Strains of Influenza Disease, for Groups Who Received the Booster Dose at Month 12
Description: A seroprotected subject was defined as a vaccinated subject with serum Hemagglutination Inhibition (HI) titer ≥ 1:40. The 2 flu strains assessed were A/Vietnam/1194/2004 (H5N1) and A/Indonesia/5/2005 (H5N1).
Time Frame: At Day 0, Day 21, Day 42, Month 6, Month 12, Month 12 + 7 Days, Month 12 + 21 Days
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/12 Group | GSK1562902A V/V/12 Group | GSK1562902A 2V/I/12 Group | GSK1562902A 2V/V/12 Group
Number analyzed (Participants) | 59 | 60 | 55 | 55
Participants
  A/Indonesia, Day 0 | 0 | 0 | 0 | 0
  A/Indonesia, Day 21: number analyzed (Participants) | 58 | 60 | 55 | 55
  A/Indonesia, Day 21 | 5 | 3 | 1 | 0
  A/Indonesia, Day 42: number analyzed (Participants) | 0 | 0 | 49 | 48
  A/Indonesia, Day 42 |  |  | 24 | 20
  A/Indonesia, Month 6: number analyzed (Participants) | 59 | 57 | 52 | 51
  A/Indonesia, Month 6 | 0 | 1 | 7 | 1
  A/Indonesia, Month 12: number analyzed (Participants) | 52 | 52 | 41 | 55
  A/Indonesia, Month 12 | 2 | 2 | 0 | 5
  A/Indonesia, Month 12 + 7 Days: number analyzed (Participants) | 50 | 51 | 40 | 43
  A/Indonesia, Month 12 + 7 Days | 40 | 44 | 34 | 39
  A/Indonesia, Month 12 + 21 Days: number analyzed (Participants) | 50 | 51 | 40 | 43
  A/Indonesia, Month 12 + 21 Days | 42 | 49 | 36 | 43
  A/Vietnam, Day 0 | 0 | 0 | 0 | 0
  A/Vietnam, Day 21: number analyzed (Participants) | 58 | 60 | 55 | 55
  A/Vietnam, Day 21 | 26 | 24 | 25 | 17
  A/Vietnam, Day 42: number analyzed (Participants) | 0 | 0 | 49 | 48
  A/Vietnam, Day 42 |  |  | 45 | 43
  A/Vietnam, Month 6: number analyzed (Participants) | 59 | 57 | 52 | 51
  A/Vietnam, Month 6 | 15 | 10 | 36 | 24
  A/Vietnam, Month 12: number analyzed (Participants) | 52 | 52 | 41 | 44
  A/Vietnam, Month 12 | 6 | 10 | 9 | 17
  A/Vietnam, Month 12 + 7 days: number analyzed (Participants) | 50 | 51 | 40 | 43
  A/Vietnam, Month 12 + 7 days | 45 | 49 | 37 | 40
  A/Vietnam, Month 12 + 21 Days: number analyzed (Participants) | 50 | 51 | 40 | 43
  A/Vietnam, Month 12 + 21 Days | 46 | 50 | 38 | 43

34. Secondary Outcome: GMTs of H5N1 HI Antibody Titers, for Groups Who Received Booster Dose at Month 6
Description: GMTs were calculated for H5N1 HI antibodies against the A/Vietnam/1194/2004 or A/Indonesia/05/2005 strains.
Time Frame: At Day 0, Day 21, Day 42, Month 6, Month 6+ 7 Days, Month 6+ 21 Days, Month 12 and at Month 18
Population: This analysis was performed on the According-to-Protocol (ATP) Cohort for Persistence, which included all evaluable subjects for whom long term immunogenicity data were available and who complied with the inclusion/exclusion criteria defined in the protocol. Day 42 data were available only from subjects who received 3 vaccine doses.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 51 | 49 | 47 | 44
Titers
  A/Indonesia, Day 0 | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  A/Indonesia, Day 21 | 6.5 [5.4 to 7.7] | 5.6 [5.1 to 6.0] | 6.3 [5.2 to 7.6] | 5.4 [5.0 to 5.8]
  A/Indonesia, Day 42: number analyzed (Participants) | 0 | 0 | 41 | 39
  A/Indonesia, Day 42 |  |  | 22.5 [14.8 to 34.3] | 16.7 [10.8 to 25.8]
  A/Indonesia, Month 6: number analyzed (Participants) | 50 | 44 | 46 | 44
  A/Indonesia, Month 6 | 5.5 [5.0 to 6.1] | 5.3 [4.9 to 5.7] | 8.5 [6.4 to 11.2] | 7.0 [5.8 to 8.4]
  A/Indonesia, Month 6 + 7 Days: number analyzed (Participants) | 48 | 42 | 45 | 42
  A/Indonesia, Month 6 + 7 Days | 142.6 [102.7 to 197.9] | 64.5 [40.1 to 103.7] | 124.1 [75.2 to 204.8] | 59.9 [38.1 to 94.3]
  A/Indonesia, Month 6 + 21 Days: number analyzed (Participants) | 47 | 43 | 46 | 42
  A/Indonesia, Month 6 + 21 Days | 290.8 [202.1 to 418.3] | 97.9 [63.3 to 151.2] | 383.5 [245.2 to 599.7] | 120.9 [76.9 to 190.1]
  A/Indonesia, Month 12: number analyzed (Participants) | 45 | 43 | 45 | 42
  A/Indonesia, Month 12 | 44.6 [28.6 to 69.5] | 17.6 [11.8 to 26.2] | 56.6 [33.7 to 95.0] | 23.8 [14.5 to 38.9]
  A/Indonesia, Month 18: number analyzed (Participants) | 44 | 42 | 46 | 40
  A/Indonesia, Month 18 | 31.1 [20.3 to 47.5] | 19.8 [13.3 to 29.7] | 50.6 [32.0 to 79.9] | 28.3 [17.0 to 47.0]
  A/Vietnam, Day 0 | 5.0 [5.0 to 5.0] | 5.2 [5.2 to 5.6] | 5.2 [4.8 to 5.7] | 5.8 [4.7 to 7.2]
  A/Vietnam, Day 21 | 20.7 [13.9 to 30.7] | 15.8 [10.9 to 23.0] | 34.3 [21.4 to 55.0] | 30.8 [18.2 to 52.2]
  A/Vietnam, Day 42: number analyzed (Participants) | 0 | 0 | 41 | 39
  A/Vietnam, Day 42 |  |  | 220.6 [145.4 to 334.6] | 275.1 [178.2 to 424.7]
  A/Vietnam, Month 6: number analyzed (Participants) | 50 | 44 | 46 | 44
  A/Vietnam, Month 6 | 11.6 [8.6 to 15.5] | 9.7 [7.3 to 12.9] | 29.6 [19.7 to 44.4] | 31.3 [20.2 to 48.5]
  A/Vietnam, Month 6 + 7 Days: number analyzed (Participants) | 48 | 42 | 45 | 42
  A/Vietnam, Month 6 + 7 Days | 209.0 [152.7 to 286.2] | 215.4 [137.8 to 336.6] | 191.0 [117.3 to 311.0] | 211.7 [133.0 to 337.0]
  A/Vietnam, Month 6 + 21 Days: number analyzed (Participants) | 47 | 43 | 46 | 42
  A/Vietnam, Month 6 + 21 Days | 411.1 [291.3 to 580.3] | 317.4 [197.5 to 510.1] | 542.1 [340.8 to 862.5] | 359.2 [220.2 to 585.9]
  A/Vietnam, Month 12: number analyzed (Participants) | 45 | 43 | 45 | 42
  A/Vietnam, Month 12 | 66.0 [43.0 to 101.1] | 63.8 [40.6 to 100.3] | 107.1 [66.4 to 172.8] | 101.6 [62.4 to 165.3]
  A/Vietnam, Month 18: number analyzed (Participants) | 44 | 42 | 46 | 40
  A/Vietnam, Month 18 | 24.3 [16.3 to 36.4] | 25.7 [16.3 to 40.4] | 45.1 [28.8 to 70.7] | 46.4 [27.7 to 77.7]

35. Secondary Outcome: Number of Seroconverted Subjects for H5N1 HI Antibodies Against 2 Strains of Influenza Disease, for Groups Who Received Booster Dose at Month 6
Description: A seroconverted (SCR) subject was defined as a vaccinated subject who had either a pre-vaccination titer <1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and at least a four-fold increase in post-vaccination titer. The 2 flu strains assessed were A/Vietnam/1194/2004 (H5N1) and A/Indonesia/5/2005 (H5N1).
Time Frame: At Day 21, Day 42, Month 6, Month 6 + 7 Days, Month 6 + 21 Days, Month 12 and Month 18
Population: This analysis was performed on the ATP Cohort for Immunogenicity and ATP Cohort for Persistence (only for M6+D7/D21, M18), which included all evaluable subjects for whom immunogenicity data were available and who complied with the criteria defined in the protocol. Day 42 data were available only from subjects who received 3 vaccine doses.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 50 | 53 | 46 | 49
Participants
  A/Indonesia, Day 21: number analyzed (Participants) | 50 | 53 | 45 | 49
  A/Indonesia, Day 21 | 0 | 3 | 0 | 3
  A/Indonesia, Day 42: number analyzed (Participants) | 0 | 0 | 39 | 43
  A/Indonesia, Day 42 |  |  | 15 | 23
  A/Indonesia, Month 6: number analyzed (Participants) | 45 | 52 | 45 | 48
  A/Indonesia, Month 6 | 0 | 0 | 2 | 4
  A/Indonesia, Month 6 + 7 Days: number analyzed (Participants) | 48 | 42 | 45 | 42
  A/Indonesia, Month 6 + 7 Days | 43 | 31 | 38 | 28
  A/Indonesia, Month 6 + 21 Days: number analyzed (Participants) | 47 | 43 | 46 | 42
  A/Indonesia, Month 6 + 21 Days | 46 | 35 | 42 | 35
  A/Indonesia, Month 12: number analyzed (Participants) | 43 | 47 | 43 | 46
  A/Indonesia, Month 12 | 16 | 29 | 19 | 31
  A/Indonesia, Month 18: number analyzed (Participants) | 44 | 42 | 46 | 40
  A/Indonesia, Month 18 | 26 | 18 | 28 | 20
  A/Vietnam, Day 21: number analyzed (Participants) | 50 | 53 | 45 | 49
  A/Vietnam, Day 21 | 19 | 24 | 23 | 29
  A/Vietnam, Day 42: number analyzed (Participants) | 0 | 0 | 39 | 43
  A/Vietnam, Day 42 |  |  | 36 | 40
  A/Vietnam, Month 6: number analyzed (Participants) | 45 | 52 | 45 | 48
  A/Vietnam, Month 6 | 5 | 13 | 25 | 25
  A/Vietnam, Month 6 + 7 Days: number analyzed (Participants) | 48 | 42 | 45 | 42
  A/Vietnam, Month 6 + 7 Days | 43 | 36 | 29 | 27
  A/Vietnam, Month 6 + 21 Days: number analyzed (Participants) | 47 | 43 | 46 | 42
  A/Vietnam, Month 6 + 21 Days | 46 | 38 | 41 | 34
  A/Vietnam, Month 12: number analyzed (Participants) | 43 | 47 | 43 | 46
  A/Vietnam, Month 12 | 33 | 35 | 32 | 37
  A/Vietnam, Month 18: number analyzed (Participants) | 44 | 42 | 46 | 40
  A/Vietnam, Month 18 | 11 | 15 | 9 | 7

36. Secondary Outcome: Seroconversion Factor for H5N1 HI Antibodies Against 2 Strains of Influenza Disease, for Groups Who Received the Booster Dose at Month 6
Description: The seroconversion factor (SCF) was defined as the fold change in serum hemagglutination inhibition (HI) geometric mean titers (GMTs) post vaccination compared to Day 0. The 2 flu strains assessed were A/Vietnam/1194/2004 (H5N1) and A/Indonesia/5/2005 (H5N1).
Time Frame: At Day 21, Day 42, Month 6, Month 6 + 7 Days, Month 6 + 21 Days, Month 12 and Month 18
Population: as for outcome 35
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Increase
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 66 | 63 | 61 | 64
Fold Increase
  A/Indonesia, Day 21 | 1.1 [1.0 to 1.2] | 1.3 [1.1 to 1.5] | 1.1 [1.0 to 1.3] | 1.2 [1.0 to 1.4]
  A/Indonesia, Day 42: number analyzed (Participants) | 0 | 0 | 52 | 54
  A/Indonesia, Day 42 |  |  | 4.1 [2.8 to 6.0] | 4.6 [3.2 to 6.8]
  A/Indonesia, Month 6: number analyzed (Participants) | 60 | 60 | 61 | 63
  A/Indonesia, Month 6 | 1.0 [1.0 to 1.1] | 1.1 [1.0 to 1.3] | 1.6 [1.4 to 2.0] | 1.6 [1.3 to 2.0]
  A/Indonesia, Month 6 + 7 Days: number analyzed (Participants) | 48 | 42 | 45 | 42
  A/Indonesia, Month 6 + 7 Days | 25.8 [18.5 to 36.0] | 12.2 [7.6 to 19.6] | 14.9 [8.6 to 26.0] | 8.6 [5.6 to 13.2]
  A/Indonesia, Month 6 + 21 Days: number analyzed (Participants) | 47 | 43 | 46 | 42
  A/Indonesia, Month 6 + 21 Days | 52.5 [36.7 to 75.0] | 18.5 [11.9 to 28.8] | 45.3 [29.9 to 68.5] | 17.5 [11.2 to 27.4]
  A/Indonesia, Month 12: number analyzed (Participants) | 58 | 54 | 56 | 60
  A/Indonesia, Month 12 | 2.9 [2.1 to 4.0] | 8.9 [5.8 to 13.6] | 5.5 [3.7 to 8.3] | 11.6 [7.4 to 18.2]
  A/Indonesia, Month 18: number analyzed (Participants) | 44 | 42 | 46 | 40
  A/Indonesia, Month 18 | 5.7 [3.7 to 8.5] | 3.7 [2.5 to 5.7] | 6.0 [4.0 to 9.0] | 4.3 [2.7 to 6.7]
  A/Vietnam, Day 21 | 3.0 [2.2 to 4.0] | 4.0 [2.8 to 5.8] | 5.7 [3.8 to 8.5] | 5.4 [3.8 to 7.9]
  A/Vietnam, Day 42: number analyzed (Participants) | 0 | 0 | 52 | 54
  A/Vietnam, Day 42 |  |  | 50.3 [34.8 to 72.7] | 40.8 [27.5 to 60.5]
  A/Vietnam, Month 6: number analyzed (Participants) | 60 | 60 | 61 | 63
  A/Vietnam, Month 6 | 1.7 [1.4 to 2.1] | 2.4 [1.8 to 3.2] | 6.4 [4.5 to 8.9] | 6.0 [4.3 to 8.5]
  A/Vietnam, Month 6 + 7 Days: number analyzed (Participants) | 48 | 42 | 45 | 42
  A/Vietnam, Month 6 + 7 Days | 17.5 [12.1 to 25.1] | 21.6 [13.1 to 35.5] | 6.5 [4.1 to 10.4] | 6.6 [4.1 to 10.6]
  A/Vietnam, Month 6 + 21 Days: number analyzed (Participants) | 47 | 43 | 46 | 42
  A/Vietnam, Month 6 + 21 Days | 34.7 [23.9 to 50.5] | 32.3 [19.8 to 52.7] | 18.3 [11.6 to 28.9] | 11.0 [6.8 to 17.9]
  A/Vietnam, Month 12: number analyzed (Participants) | 58 | 54 | 56 | 60
  A/Vietnam, Month 12 | 9.6 [6.3 to 14.7] | 14.3 [9.6 to 21.4] | 19.0 [12.9 to 28.1] | 22.5 [14.5 to 34.9]
  A/Vietnam, Month 18: number analyzed (Participants) | 44 | 42 | 46 | 40
  A/Vietnam, Month 18 | 2.1 [1.5 to 3.1] | 2.7 [1.7 to 4.2] | 1.5 [1.1 to 2.2] | 1.5 [0.9 to 2.3]

37. Secondary Outcome: Number of Seroprotected Subjects for H5N1 HI Antibodies Against 2 Strains of Influenza Disease, for Groups Who Received Booster Dose at Month 6
Description: A seroprotected (SPR) subject was defined as a vaccinated subject with serum Hemagglutination Inhibition (HI) titer ≥ 1:40. The 2 flu strains assessed were A/Vietnam/1194/2004 (H5N1) and A/Indonesia/5/2005 (H5N1).
Time Frame: At Day 0, Day 21, Day 42, Month 6, Month 6+ 7 Days, Month 6+ 21 Days, Month 12 and Month 18
Population: This analysis was performed on the ATP Cohort for Immunogenicity and ATP Cohort for Persistence (only for M18), which included all evaluable subjects for whom immunogenicity data were available and who complied with the inclusion/exclusion criteria defined in the protocol. Day 42 data were available only from subjects who received 3 vaccine doses.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 50 | 53 | 46 | 49
Participants
  A/Indonesia, Day 0: number analyzed (Participants) | 50 | 53 | 45 | 49
  A/Indonesia, Day 0 | 0 | 0 | 0 | 0
  A/Indonesia, Day 21: number analyzed (Participants) | 50 | 53 | 45 | 49
  A/Indonesia, Day 21 | 0 | 3 | 0 | 3
  A/Indonesia, Day 42: number analyzed (Participants) | 0 | 0 | 39 | 43
  A/Indonesia, Day 42 |  |  | 15 | 23
  A/Indonesia, Month 6: number analyzed (Participants) | 45 | 52 | 45 | 48
  A/Indonesia, Month 6 | 0 | 0 | 2 | 4
  A/Indonesia, Month 6 + 7 Days: number analyzed (Participants) | 43 | 50 | 43 | 47
  A/Indonesia, Month 6 + 7 Days | 32 | 46 | 31 | 40
  A/Indonesia, Month 6 + 21 Days: number analyzed (Participants) | 44 | 49 | 43 | 48
  A/Indonesia, Month 6 + 21 Days | 37 | 48 | 37 | 45
  A/Indonesia, Month 12: number analyzed (Participants) | 43 | 47 | 43 | 46
  A/Indonesia, Month 12 | 16 | 29 | 19 | 31
  A/Indonesia, Month 18: number analyzed (Participants) | 44 | 42 | 46 | 40
  A/Indonesia, Month 18 | 26 | 18 | 30 | 21
  A/Vietnam, Day 0: number analyzed (Participants) | 50 | 53 | 45 | 49
  A/Vietnam, Day 0 | 0 | 0 | 2 | 1
  A/Vietnam, Day 21: number analyzed (Participants) | 50 | 53 | 45 | 49
  A/Vietnam, Day 21 | 19 | 24 | 24 | 29
  A/Vietnam, Day 42: number analyzed (Participants) | 0 | 0 | 39 | 43
  A/Vietnam, Day 42 |  |  | 36 | 40
  A/Vietnam, Month 6: number analyzed (Participants) | 45 | 52 | 45 | 48
  A/Vietnam, Month 6 | 6 | 13 | 26 | 25
  A/Vietnam, Month 6 + 7 Days: number analyzed (Participants) | 43 | 50 | 43 | 47
  A/Vietnam, Month 6 + 7 Days | 39 | 49 | 38 | 42
  A/Vietnam, Month 6 + 21 Days: number analyzed (Participants) | 44 | 49 | 43 | 48
  A/Vietnam, Month 6 + 21 Days | 40 | 48 | 39 | 45
  A/Vietnam, Month 12: number analyzed (Participants) | 43 | 47 | 43 | 46
  A/Vietnam, Month 12 | 33 | 35 | 33 | 37
  A/Vietnam, Month 18: number analyzed (Participants) | 44 | 42 | 46 | 40
  A/Vietnam, Month 18 | 21 | 24 | 30 | 24

38. Secondary Outcome: Number of Booster Seroconverted Subjects Against 2 Strains of Influenza Disease, A/Vietnam/1194/2004 and A/Indonesia/5/2005, for Groups Who Received Booster Dose at Month 12
Description: Booster seroconversion (SCR) was defined as: For seronegative subjects at pre-booster (Month 12), antibody titer ≥ 1:40 at Month 12 + 7 days; For seropositive subjects at pre-booster (Month 12), antibody titer at Month 12 + 7 days ≥ 4 fold the pre-vaccination antibody titer at Month 12.
Time Frame: At Month 12 + 7 Days, Month 12 + 21 Days and Month 18
Population: This analysis was performed on the ATP Cohort for Immunogenicity and ATP Cohort for Persistence (only for M18), which included all evaluable subjects for whom immunogenicity data/long term immunogenicity data were available and who complied with the inclusion/exclusion criteria as defined in the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/12 Group | GSK1562902A V/V/12 Group | GSK1562902A 2V/I/12 Group | GSK1562902A 2V/V/12 Group
Number analyzed (Participants) | 50 | 51 | 40 | 43
Participants
  A/Indonesia, Month 12 + 7 Days | 38 | 43 | 34 | 39
  A/Indonesia, Month 12 + 21 Days | 41 | 49 | 36 | 43
  A/Indonesia, Month 18: number analyzed (Participants) | 44 | 48 | 39 | 40
  A/Indonesia, Month 18 | 39 | 34 | 37 | 34
  A/Vietnam, Month 12 + 7 Days | 43 | 46 | 34 | 38
  A/Vietnam, Month 12 + 21 Days | 44 | 50 | 37 | 43
  A/Vietnam, Month 18: number analyzed (Participants) | 44 | 48 | 39 | 40
  A/Vietnam, Month 18 | 30 | 33 | 34 | 29

39. Secondary Outcome: Booster Factor of H5N1 HI Antibodies Against 2 Strains of Influenza Disease, for Groups Who Received Booster Dose at Month 12
Description: Booster Factor (Seroconversion Factor booster) was defined as the fold change in H5N1 HI antibodies between the pre- and post-booster vaccination time-points (mean[log10(POST/M12)]). The 2 flu strains assessed were A/Vietnam/1194/2004 and A/Indonesia/05/2005, for groups who received the booster dose at Month 12.
Time Frame: At Month 12 + 7 Days and at Month 12 + 21 Days
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Increase
Arm/Group | GSK1562902A V/I/12 Group | GSK1562902A V/V/12 Group | GSK1562902A 2V/I/12 Group | GSK1562902A 2V/V/12 Group
Number analyzed (Participants) | 51 | 50 | 43 | 40
Fold Increase
  A/Indonesia, Month 12 + 7 Days | 33.1 [21.3 to 51.6] | 16.7 [11.3 to 24.7] | 29.1 [17.0 to 49.6] | 18.7 [11.7 to 29.9]
  A/Indonesia, Month 12 + 21 Days | 70.9 [47.0 to 107.0] | 23.8 [15.7 to 35.9] | 75.8 [54.2 to 106.1] | 33.7 [21.0 to 54.1]
  A/Vietnam, Month 12 + 7 Days | 35.2 [22.4 to 55.3] | 27.5 [17.4 to 43.5] | 21.9 [12.7 to 37.9] | 17.6 [10.8 to 28.8]
  A/Vietnam, Month 12 + 21 Days | 65.8 [42.2 to 102.6] | 41.1 [25.8 to 65.4] | 57.6 [38.6 to 86.1] | 30.2 [18.6 to 48.8]

40. Secondary Outcome: Booster Factor of H5N1 HI Antibodies Against 2 Strains of Influenza Disease, for Groups Who Received Booster Dose at Month 12
Description: as for outcome 39
Time Frame: At Month 12 + 7 Days, Month 12 + 21 Days and at Month 18
Population: The analysis was performed on the ATP Cohort for persistence, which included all evaluable subjects for whom long term immunogenicity data were available and who complied with the inclusion/exclusion criteria as defined in the protocol.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Increase
Arm/Group | GSK1562902A V/I/12 Group | GSK1562902A V/V/12 Group | GSK1562902A 2V/I/12 Group | GSK1562902A 2V/V/12 Group
Number analyzed (Participants) | 47 | 48 | 40 | 40
Fold Increase
  A/Indonesia, Month 12 + 7 Days | 35.2 [22.4 to 55.4] | 16.8 [11.2 to 25.2] | 27.9 [15.8 to 49.2] | 18.7 [11.7 to 29.9]
  A/Indonesia, Month 12 + 21 Days | 78.7 [52.9 to 117.2] | 23.6 [15.4 to 36.3] | 76.2 [53.2 to 109.0] | 33.7 [21.0 to 54.1]
  A/Indonesia, Month 18: number analyzed (Participants) | 44 | 48 | 39 | 40
  A/Indonesia, Month 18 | 25.1 [15.8 to 39.8] | 10.3 [6.6 to 16.0] | 44.5 [27.9 to 71.0] | 21.3 [13.2 to 34.4]
  A/Vietnam, Month 12 + 7 Days | 37.9 [24.0 to 59.8] | 28.9 [18.1 to 46.3] | 19.9 [11.2 to 35.3] | 17.6 [10.8 to 28.8]
  A/Vietnam, Month 12 + 21 Days | 73.6 [47.9 to 113.3] | 43.1 [26.6 to 69.6] | 55.7 [36.4 to 85.3] | 30.2 [18.6 to 48.8]
  A/Vietnam, Month 18: number analyzed (Participants) | 44 | 48 | 39 | 40
  A/Vietnam, Month 18 | 12.0 [7.3 to 19.8] | 10.2 [6.4 to 16.1] | 18.6 [11.1 to 31.2] | 10.2 [6.2 to 16.8]

41. Secondary Outcome: Frequency of Influenza-specific CD4/CD8 T-cells (Per 10E6 T-cells) in Tests Identified as Producing at Least Two Out of Four Different Cytokines, for Groups Who Received Booster Dose at Month 6
Description: Among cytokines expressed after background reduction were cluster of differentiation 4 all doubles (CD4 All Doubles), cluster of differentiation 40-ligand (CD40-L), interleukin-2 (IL-2), interferon-gamma (IFN-γ) and tumour necrosis factor-alpha (TNF-α). The 2 flu strains assessed were A/Indonesia/05/2005 and A/Vietnam/1194/2004.
Time Frame: At Day 0, Month 6, Month 6 + 7 Days, Month 6 + 21 Days, Month 12 and Month 18
Population: This analysis was performed on the ATP Cohort for Immunogenicity and ATP Cohort for Persistence (only for M12, M18), which included all evaluable subjects for whom immunogenicity data were available and who complied with the inclusion/exclusion criteria as defined in the protocol.
Measure: Mean (Standard Deviation); unit: cells/million T-cells
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 41 | 42 | 36 | 35
cells/million T-cells
  CD4 All Doubles - A/Vietnam, Day 0 | 412.03 (487.53) | 467.30 (333.87) | 395.60 (477.64) | 469.25 (470.89)
  CD4 All Doubles - A/Vietnam, Month 6: number analyzed (Participants) | 30 | 32 | 32 | 27
  CD4 All Doubles - A/Vietnam, Month 6 | 600.07 (901.78) | 807.14 (806.63) | 896.67 (627.38) | 1071.19 (923.45)
  CD4 All Doubles - A/Vietnam, Month 6 + 7 Days: number analyzed (Participants) | 29 | 26 | 21 | 22
  CD4 All Doubles - A/Vietnam, Month 6 + 7 Days | 1120.95 (2182.54) | 1369.15 (1224.75) | 1914.50 (1757.90) | 1769.33 (1024.50)
  CD4 All Doubles - A/Vietnam, Month 6 + 21 Days: number analyzed (Participants) | 32 | 30 | 25 | 31
  CD4 All Doubles - A/Vietnam, Month 6 + 21 Days | 1619.46 (1899.48) | 1531.69 (1741.38) | 1489.30 (1564.28) | 1953.30 (2219.16)
  CD4 All Doubles - A/Indonesia, Month 12: number analyzed (Participants) | 33 | 33 | 35 | 31
  CD4 All Doubles - A/Indonesia, Month 12 | 1196.05 (1279.60) | 1461.46 (1972.69) | 1512.82 (996.79) | 1243.41 (1434.39)
  CD4 All Doubles - A/Vietnam, Month 12: number analyzed (Participants) | 33 | 33 | 35 | 31
  CD4 All Doubles - A/Vietnam, Month 12 | 1316.68 (1359.39) | 1431.92 (1291.80) | 1506.94 (1086.61) | 1220.87 (2280.45)
  CD4 All Doubles - A/Indonesia, Month 18: number analyzed (Participants) | 37 | 36 | 33 | 34
  CD4 All Doubles - A/Indonesia, Month 18 | 1192.82 (1000.13) | 1767.82 (1194.85) | 1978.73 (1138.17) | 1550.40 (1557.30)
  CD4 All Doubles - A/Vietnam, Month 18: number analyzed (Participants) | 37 | 36 | 33 | 34
  CD4 All Doubles - A/Vietnam, Month 18 | 1194.69 (1073.65) | 1790.56 (1178.39) | 1676.20 (1267.85) | 1560.54 (1546.70)
  CD4 CD40L - A/Vietnam, Day 0 | 350.86 (455.52) | 446.27 (318.18) | 387.68 (458.40) | 441.16 (460.09)
  CD4 CD40L - A/Vietnam, Month 6: number analyzed (Participants) | 30 | 32 | 32 | 27
  CD4 CD40L - A/Vietnam, Month 6 | 593.74 (885.01) | 809.47 (777.20) | 867.92 (591.04) | 1046.99 (893.54)
  CD4 CD40L - A/Vietnam, Month 6 + 7 Days: number analyzed (Participants) | 29 | 26 | 21 | 22
  CD4 CD40L - A/Vietnam, Month 6 + 7 Days | 1084.46 (2123.12) | 1298.95 (1153.28) | 1818.39 (1603.64) | 1717.69 (990.51)
  CD4 CD40L - A/Vietnam, Month 6 + 21 Days: number analyzed (Participants) | 32 | 30 | 25 | 31
  CD4 CD40L - A/Vietnam, Month 6 + 21 Days | 1588.60 (1855.12) | 1487.73 (1663.98) | 1480.21 (1520.92) | 1880.07 (2151.87)
  CD4 CD40L - A/Indonesia, Month 12: number analyzed (Participants) | 33 | 33 | 35 | 31
  CD4 CD40L - A/Indonesia, Month 12 | 1183.85 (1255.59) | 1448.44 (1973.98) | 1505.73 (985.99) | 1221.20 (1371.18)
  CD4 CD40L - A/Vietnam, Month 12: number analyzed (Participants) | 33 | 33 | 35 | 31
  CD4 CD40L - A/Vietnam, Month 12 | 1238.24 (1362.58) | 1390.02 (1288.92) | 1474.26 (1073.10) | 1152.29 (2263.92)
  CD4 CD40L - A/Indonesia, Month 18: number analyzed (Participants) | 37 | 36 | 33 | 34
  CD4 CD40L - A/Indonesia, Month 18 | 1172.36 (985.13) | 1747.96 (1151.98) | 1975.69 (1126.07) | 1522.12 (1553.48)
  CD4 CD40L- A/Vietnam, Month 18: number analyzed (Participants) | 37 | 36 | 33 | 34
  CD4 CD40L- A/Vietnam, Month 18 | 1162.79 (1043.15) | 1738.30 (1140.59) | 1640.12 (1252.01) | 1518.75 (1489.22)
  CD4 IL-2 - A/Vietnam, Day 0 | 262.64 (339.55) | 264.51 (249.40) | 230.40 (360.46) | 289.83 (385.44)
  CD4 IL-2 - A/Vietnam, Month 6: number analyzed (Participants) | 30 | 32 | 32 | 27
  CD4 IL-2 - A/Vietnam, Month 6 | 450.20 (815.29) | 601.02 (736.05) | 648.07 (584.83) | 719.07 (763.89)
  CD4 IL-2 - A/Vietnam, Month 6 + 7 Days: number analyzed (Participants) | 29 | 26 | 21 | 22
  CD4 IL-2 - A/Vietnam, Month 6 + 7 Days | 861.32 (1997.52) | 890.90 (1030.87) | 1390.30 (1480.20) | 1147.31 (980.42)
  CD4 IL-2 - A/Vietnam, Month 6 + 21 Days: number analyzed (Participants) | 32 | 30 | 25 | 31
  CD4 IL-2 - A/Vietnam, Month 6 + 21 Days | 1238.06 (1759.16) | 1036.73 (1545.30) | 965.41 (1302.89) | 1380.65 (1761.07)
  CD4 IL-2 - A/Indonesia, Month 12: number analyzed (Participants) | 33 | 33 | 35 | 31
  CD4 IL-2 - A/Indonesia, Month 12 | 1001.88 (1156.16) | 1169.25 (1630.99) | 1278.49 (908.04) | 1041.21 (1250.37)
  CD4 IL-2 - A/Vietnam, Month 12: number analyzed (Participants) | 33 | 33 | 35 | 31
  CD4 IL-2 - A/Vietnam, Month 12 | 1119.56 (1261.18) | 1160.06 (1049.95) | 1264.64 (1008.46) | 999.23 (2005.29)
  CD4 IL-2 - A/Indonesia, Month 18: number analyzed (Participants) | 37 | 36 | 33 | 34
  CD4 IL-2 - A/Indonesia, Month 18 | 999.22 (844.48) | 1412.43 (986.25) | 1480.68 (1040.08) | 1248.66 (1383.46)
  CD4 IL-2- A/Vietnam, Month 18: number analyzed (Participants) | 37 | 36 | 33 | 34
  CD4 IL-2- A/Vietnam, Month 18 | 1011.14 (921.27) | 1487.16 (1006.20) | 1434.59 (1156.89) | 1140.29 (1374.45)
  CD4 IFN-γ - A/Vietnam, Day 0 | 303.97 (403.90) | 267.88 (316.20) | 275.09 (299.79) | 331.35 (379.46)
  CD4 IFN-γ - A/Vietnam, Month 6: number analyzed (Participants) | 30 | 32 | 32 | 27
  CD4 IFN-γ - A/Vietnam, Month 6 | 309.94 (596.66) | 486.23 (524.58) | 406.50 (364.57) | 543.11 (607.67)
  CD4 IFN-γ - A/Vietnam, Month 6 + 7 Days: number analyzed (Participants) | 29 | 26 | 21 | 22
  CD4 IFN-γ - A/Vietnam, Month 6 + 7 Days | 632.73 (848.00) | 683.35 (702.66) | 826.27 (856.63) | 887.74 (412.30)
  CD4 IFN-γ - A/Vietnam, Month 6 + 21 Days: number analyzed (Participants) | 32 | 30 | 25 | 31
  CD4 IFN-γ - A/Vietnam, Month 6 + 21 Days | 769.33 (858.31) | 831.31 (964.67) | 712.10 (806.47) | 908.75 (952.74)
  CD4 IFN-γ - A/Indonesia, Month 12: number analyzed (Participants) | 33 | 33 | 35 | 31
  CD4 IFN-γ - A/Indonesia, Month 12 | 615.47 (624.58) | 829.05 (903.32) | 752.50 (525.81) | 746.33 (727.94)
  CD4 IFN-γ - A/Vietnam, Month 12: number analyzed (Participants) | 33 | 33 | 35 | 31
  CD4 IFN-γ - A/Vietnam, Month 12 | 751.16 (604.70) | 851.71 (727.68) | 817.48 (568.54) | 832.49 (1138.08)
  CD4 IFN-γ - A/Indonesia, Month 18: number analyzed (Participants) | 37 | 36 | 33 | 34
  CD4 IFN-γ - A/Indonesia, Month 18 | 657.19 (622.98) | 972.81 (1026.12) | 1017.82 (655.54) | 883.75 (969.20)
  CD4 IFN-γ - A/Vietnam, Month 18: number analyzed (Participants) | 37 | 36 | 33 | 34
  CD4 IFN-γ - A/Vietnam, Month 18 | 698.55 (804.64) | 1018.23 (959.34) | 1066.89 (845.76) | 949.06 (949.59)
  CD4 TNF-α - A/Vietnam, Day 0 | 213.17 (314.89) | 290.55 (244.57) | 248.53 (334.40) | 262.12 (309.11)
  CD4 TNF-α - A/Vietnam, Month 6: number analyzed (Participants) | 30 | 32 | 32 | 27
  CD4 TNF-α - A/Vietnam, Month 6 | 389.55 (823.34) | 459.89 (709.54) | 501.89 (496.82) | 684.19 (700.61)
  CD4 TNF-α - A/Vietnam, Month 6 + 7 Days: number analyzed (Participants) | 29 | 26 | 21 | 22
  CD4 TNF-α - A/Vietnam, Month 6 + 7 Days | 605.80 (1282.37) | 700.69 (893.07) | 1160.60 (1524.45) | 972.71 (668.12)
  CD4 TNF-α - A/Vietnam, Month 6 + 21 Days: number analyzed (Participants) | 32 | 30 | 25 | 31
  CD4 TNF-α - A/Vietnam, Month 6 + 21 Days | 880.12 (1327.15) | 971.44 (1419.68) | 881.65 (1218.69) | 1227.63 (1871.42)
  CD4 TNF-α - A/Indonesia, Month 12: number analyzed (Participants) | 33 | 33 | 35 | 31
  CD4 TNF-α - A/Indonesia, Month 12 | 914.94 (1053.34) | 1125.16 (1559.54) | 1235.28 (813.44) | 1148.53 (1208.96)
  CD4 TNF-α - A/Vietnam, Month 12: number analyzed (Participants) | 33 | 33 | 35 | 31
  CD4 TNF-α - A/Vietnam, Month 12 | 970.90 (1091.23) | 1047.93 (978.11) | 1238.05 (858.40) | 1096.87 (1906.75)
  CD4 TNF-α - A/Indonesia, Month 18: number analyzed (Participants) | 37 | 36 | 33 | 34
  CD4 TNF-α - A/Indonesia, Month 18 | 922.42 (794.83) | 1318.59 (923.86) | 1647.61 (927.11) | 1224.50 (1267.20)
  CD4 TNF-α - A/Vietnam, Month 18: number analyzed (Participants) | 37 | 36 | 33 | 34
  CD4 TNF-α - A/Vietnam, Month 18 | 877.90 (810.80) | 1314.99 (846.99) | 1232.41 (1079.43) | 1147.21 (1402.58)
  CD8 All Doubles - A/Vietnam, Day 0: number analyzed (Participants) | 41 | 40 | 36 | 34
  CD8 All Doubles - A/Vietnam, Day 0 | 67.13 (366.43) | 26.91 (128.98) | 30.44 (219.02) | 45.07 (377.44)
  CD8 All Doubles - A/Vietnam, Month 6: number analyzed (Participants) | 29 | 31 | 32 | 27
  CD8 All Doubles - A/Vietnam, Month 6 | 20.86 (222.56) | 18.86 (271.65) | 37.69 (271.61) | 40.43 (148.42)
  CD8 All Doubles - A/Vietnam, Month 6 + 7 Days: number analyzed (Participants) | 29 | 25 | 21 | 22
  CD8 All Doubles - A/Vietnam, Month 6 + 7 Days | 23.01 (290.71) | 27.73 (93.80) | 38.78 (211.71) | 32.56 (150.48)
  CD8 All Doubles - A/Vietnam, Month 6 + 21 Days: number analyzed (Participants) | 31 | 28 | 25 | 31
  CD8 All Doubles - A/Vietnam, Month 6 + 21 Days | 29.21 (281.87) | 52.59 (159.49) | 36.47 (171.22) | 16.93 (105.56)
  CD8 All Doubles - A/Indonesia, Month 12: number analyzed (Participants) | 32 | 32 | 35 | 31
  CD8 All Doubles - A/Indonesia, Month 12 | 47.78 (1206.89) | 31.69 (1136.66) | 64.08 (1893.94) | 36.18 (1567.28)
  CD8 All Doubles - A/Vietnam, Month 12: number analyzed (Participants) | 31 | 32 | 35 | 29
  CD8 All Doubles - A/Vietnam, Month 12 | 15.04 (544.79) | 21.08 (635.65) | 37.32 (744.75) | 14.09 (771.65)
  CD8 All Doubles - A/Indonesia, Month 18: number analyzed (Participants) | 37 | 35 | 33 | 33
  CD8 All Doubles - A/Indonesia, Month 18 | 48.27 (1109.56) | 24.19 (1162.30) | 82.90 (1266.82) | 34.07 (1414.34)
  CD8 All Doubles - A/Vietnam, Month 18: number analyzed (Participants) | 36 | 35 | 33 | 32
  CD8 All Doubles - A/Vietnam, Month 18 | 33.20 (623.81) | 12.14 (907.62) | 29.83 (673.80) | 11.17 (676.65)
  CD8 CD40L - A/Vietnam, Day 0: number analyzed (Participants) | 41 | 40 | 36 | 34
  CD8 CD40L - A/Vietnam, Day 0 | 7.17 (84.29) | 4.74 (71.68) | 5.49 (39.03) | 6.15 (165.75)
  CD8 CD40L - A/Vietnam, Month 6: number analyzed (Participants) | 29 | 31 | 32 | 27
  CD8 CD40L - A/Vietnam, Month 6 | 3.12 (35.61) | 7.18 (39.67) | 5.01 (69.22) | 4.81 (49.19)
  CD8 CD40L - A/Vietnam, Month 6 + 7 Days: number analyzed (Participants) | 29 | 25 | 21 | 22
  CD8 CD40L - A/Vietnam, Month 6 + 7 Days | 6.26 (71.82) | 3.55 (30.06) | 6.28 (34.99) | 5.92 (45.82)
  CD8 CD40L - A/Vietnam, Month 6 + 21 Days: number analyzed (Participants) | 31 | 28 | 25 | 31
  CD8 CD40L - A/Vietnam, Month 6 + 21 Days | 2.11 (22.77) | 4.88 (37.26) | 3.78 (33.23) | 3.21 (30.61)
  CD8 CD40L - A/Indonesia, Month 12: number analyzed (Participants) | 32 | 32 | 35 | 31
  CD8 CD40L - A/Indonesia, Month 12 | 3.92 (58.33) | 5.74 (93.30) | 9.05 (186.92) | 7.74 (144.04)
  CD8 CD40L - A/Vietnam, Month 12: number analyzed (Participants) | 31 | 32 | 35 | 29
  CD8 CD40L - A/Vietnam, Month 12 | 2.27 (33.81) | 3.40 (67.73) | 5.10 (65.14) | 3.35 (47.52)
  CD8 CD40L - A/Indonesia, Month 18: number analyzed (Participants) | 37 | 35 | 33 | 33
  CD8 CD40L - A/Indonesia, Month 18 | 5.88 (71.14) | 5.23 (269.38) | 5.25 (71.46) | 3.66 (56.08)
  CD8 CD40L - A/Vietnam, Month 18: number analyzed (Participants) | 36 | 35 | 33 | 32
  CD8 CD40L - A/Vietnam, Month 18 | 5.71 (53.55) | 2.75 (96.74) | 4.14 (95.17) | 3.07 (40.00)
  CD8 IL-2 - A/Vietnam, Day 0: number analyzed (Participants) | 41 | 40 | 36 | 34
  CD8 IL-2 - A/Vietnam, Day 0 | 36.92 (229.00) | 14.67 (100.62) | 16.98 (130.69) | 27.00 (258.14)
  CD8 IL-2 - A/Vietnam, Month 6: number analyzed (Participants) | 29 | 42 | 32 | 27
  CD8 IL-2 - A/Vietnam, Month 6 | 12.84 (129.21) | 12.58 (239.74) | 22.68 (113.81) | 25.91 (102.37)
  CD8 IL-2 - A/Vietnam, Month 6 + 7 Days: number analyzed (Participants) | 29 | 25 | 21 | 22
  CD8 IL-2 - A/Vietnam, Month 6 + 7 Days | 16.03 (218.16) | 17.04 (92.98) | 32.94 (154.53) | 26.46 (113.81)
  CD8 IL-2 - A/Vietnam, Month 6 + 21 Days: number analyzed (Participants) | 31 | 28 | 25 | 31
  CD8 IL-2 - A/Vietnam, Month 6 + 21 Days | 31.00 (185.96) | 28.04 (156.16) | 22.75 (138.13) | 13.48 (93.72)
  CD8 IL-2 - A/Indonesia, Month 12: number analyzed (Participants) | 32 | 32 | 35 | 31
  CD8 IL-2 - A/Indonesia, Month 12 | 40.26 (1211.36) | 27.79 (1135.75) | 48.91 (1897.48) | 28.61 (1566.57)
  CD8 IL-2 - A/Vietnam, Month 12: number analyzed (Participants) | 31 | 32 | 35 | 29
  CD8 IL-2 - A/Vietnam, Month 12 | 14.98 (532.13) | 21.52 (631.86) | 31.94 (746.85) | 13.31 (773.02)
  CD8 IL-2 - A/Indonesia, Month 18: number analyzed (Participants) | 37 | 35 | 33 | 33
  CD8 IL-2 - A/Indonesia, Month 18 | 43.26 (1110.98) | 19.50 (1164.40) | 66.29 (1268.66) | 33.60 (1414.79)
  CD8 IL-2 - A/Vietnam, Month 18: number analyzed (Participants) | 36 | 35 | 33 | 32
  CD8 IL-2 - A/Vietnam, Month 18 | 32.16 (615.73) | 11.75 (902.78) | 26.63 (674.63) | 9.50 (678.33)
  CD8 IFN-γ - A/Vietnam, Day 0: number analyzed (Participants) | 41 | 40 | 36 | 34
  CD8 IFN-γ - A/Vietnam, Day 0 | 29.70 (347.16) | 14.50 (125.14) | 24.17 (183.45) | 23.68 (347.01)
  CD8 IFN-γ - A/Vietnam, Month 6: number analyzed (Participants) | 29 | 31 | 32 | 27
  CD8 IFN-γ - A/Vietnam, Month 6 | 9.15 (195.76) | 15.10 (164.89) | 25.09 (269.60) | 10.92 (133.43)
  CD8 IFN-γ - A/Vietnam, Month 6 + 7 days: number analyzed (Participants) | 29 | 25 | 21 | 22
  CD8 IFN-γ - A/Vietnam, Month 6 + 7 days | 17.52 (252.30) | 6.54 (65.11) | 6.15 (190.69) | 12.90 (96.83)
  CD8 IFN-γ - A/Vietnam, Month 6 + 21 Days: number analyzed (Participants) | 31 | 28 | 25 | 31
  CD8 IFN-γ - A/Vietnam, Month 6 + 21 Days | 9.86 (272.26) | 16.87 (111.49) | 15.44 (132.81) | 11.37 (82.16)
  CD8 IFN-γ - A/Indonesia, Month 12: number analyzed (Participants) | 32 | 32 | 35 | 31
  CD8 IFN-γ - A/Indonesia, Month 12 | 3.05 (131.52) | 4.05 (147.20) | 4.11 (75.97) | 2.83 (38.52)
  CD8 IFN-γ - A/Vietnam, Month 12: number analyzed (Participants) | 31 | 32 | 35 | 29
  CD8 IFN-γ - A/Vietnam, Month 12 | 4.44 (305.15) | 4.24 (133.39) | 10.21 (83.42) | 4.42 (56.81)
  CD8 IFN-γ - A/Indonesia, Month 18: number analyzed (Participants) | 37 | 35 | 33 | 33
  CD8 IFN-γ - A/Indonesia, Month 18 | 4.74 (91.61) | 4.33 (111.98) | 4.61 (83.81) | 3.73 (97.93)
  CD8 IFN-γ - A/Vietnam, Month 18: number analyzed (Participants) | 36 | 35 | 33 | 32
  CD8 IFN-γ - A/Vietnam, Month 18 | 5.73 (64.14) | 3.55 (138.59) | 5.22 (95.47) | 3.15 (107.32)
  CD8 TNF-α - A/Vietnam, Day 0: number analyzed (Participants) | 41 | 40 | 36 | 34
  CD8 TNF-α - A/Vietnam, Day 0 | 25.46 (308.45) | 14.67 (92.23) | 22.21 (183.41) | 35.35 (219.77)
  CD8 TNF-α - A/Vietnam, Month 6: number analyzed (Participants) | 29 | 31 | 32 | 27
  CD8 TNF-α - A/Vietnam, Month 6 | 11.60 (192.99) | 17.44 (260.42) | 21.86 (254.39) | 20.44 (140.65)
  CD8 TNF-α - A/Vietnam, Month 6 + 7 Days: number analyzed (Participants) | 29 | 25 | 21 | 22
  CD8 TNF-α - A/Vietnam, Month 6 + 7 Days | 17.12 (200.81) | 14.74 (90.05) | 25.85 (186.72) | 27.99 (151.32)
  CD8 TNF-α - A/Vietnam, Month 6 + 21 Days: number analyzed (Participants) | 31 | 28 | 25 | 31
  CD8 TNF-α - A/Vietnam, Month 6 + 21 Days | 28.56 (229.92) | 38.71 (137.20) | 27.86 (156.35) | 11.99 (83.27)
  CD8 TNF-α - A/Indonesia, Month 12: number analyzed (Participants) | 32 | 32 | 35 | 31
  CD8 TNF-α - A/Indonesia, Month 12 | 46.49 (1154.66) | 27.72 (1030.52) | 57.62 (1753.76) | 31.65 (1425.49)
  CD8 TNF-α - A/Vietnam, Month 12: number analyzed (Participants) | 31 | 32 | 35 | 29
  CD8 TNF-α - A/Vietnam, Month 12 | 13.46 (423.36) | 18.89 (579.22) | 35.19 (698.32) | 12.30 (725.71)
  CD8 TNF-α - A/Indonesia, Month 18: number analyzed (Participants) | 37 | 35 | 33 | 33
  CD8 TNF-α - A/Indonesia, Month 18 | 45.67 (1033.79) | 22.55 (1002.19) | 70.09 (1200.29) | 34.37 (1369.22)
  CD8 TNF-α - A/Vietnam, Month 18: number analyzed (Participants) | 36 | 35 | 33 | 32
  CD8 TNF-α - A/Vietnam, Month 18 | 31.41 (580.62) | 12.96 (816.63) | 21.36 (614.44) | 9.31 (642.97)

42. Secondary Outcome: Frequency of Influenza-specific CD4/CD8 T-cells (Per 10E6 T-cells) in Tests Identified as Producing at Least Two Out of Four Different Cytokines, for Groups Who Received Booster Dose at Month 12
Description: as for outcome 41
Time Frame: At Day 0, Month 6, Month 12, Month 12 + 7 Days, Month 12 + 21 Days and Month 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/million T-cells
Arm/Group | GSK1562902A V/I/12 Group | GSK1562902A V/V/12 Group | GSK1562902A 2V/I/12 Group | GSK1562902A 2V/V/12 Group
Number analyzed (Participants) | 47 | 51 | 46 | 43
cells/million T-cells
  CD4 All Doubles - A/Vietnam, Day 0 | 560.41 (427.07) | 529.20 (549.34) | 542.86 (488.28) | 771.60 (788.54)
  CD4 All Doubles - A/Vietnam, Month 6: number analyzed (Participants) | 32 | 31 | 36 | 28
  CD4 All Doubles - A/Vietnam, Month 6 | 1296.63 (839.72) | 931.49 (717.72) | 1714.23 (837.39) | 1601.31 (1020.97)
  CD4 All Doubles - A/Indonesia, Month 12: number analyzed (Participants) | 33 | 34 | 23 | 31
  CD4 All Doubles - A/Indonesia, Month 12 | 1379.04 (701.03) | 1254.05 (835.74) | 1690.38 (1135.04) | 1534.37 (1256.20)
  CD4 All Doubles - A/Vietnam, Month 12: number analyzed (Participants) | 29 | 33 | 21 | 30
  CD4 All Doubles - A/Vietnam, Month 12 | 1230.51 (523.55) | 1093.54 (941.19) | 1260.93 (1118.44) | 1224.35 (2953.68)
  CD4 All Doubles - A/Indonesia, Month 12 + 7 Days: number analyzed (Participants) | 38 | 39 | 26 | 32
  CD4 All Doubles - A/Indonesia, Month 12 + 7 Days | 1979.02 (1644.97) | 1763.05 (1266.55) | 3030.85 (1974.08) | 3202.67 (7114.42)
  CD4 All Doubles - A/Vietnam, Month 12 + 7 days: number analyzed (Participants) | 41 | 40 | 26 | 33
  CD4 All Doubles - A/Vietnam, Month 12 + 7 days | 2278.65 (2822.40) | 1856.17 (1517.33) | 2953.57 (2725.45) | 3502.70 (19908.39)
  CD4 All Doubles - A/Indonesia, Month 12 + 21 Days: number analyzed (Participants) | 37 | 38 | 30 | 32
  CD4 All Doubles - A/Indonesia, Month 12 + 21 Days | 2837.94 (1587.84) | 2180.14 (2032.36) | 3600.62 (2903.90) | 3221.46 (2824.65)
  CD4 All Doubles - A/Vietnam, Month 12 + 21 Days: number analyzed (Participants) | 38 | 41 | 32 | 32
  CD4 All Doubles - A/Vietnam, Month 12 + 21 Days | 2651.19 (2181.61) | 2276.18 (1434.51) | 3386.98 (3153.08) | 3603.01 (3804.83)
  CD4 All Doubles - A/Indonesia, Month 18: number analyzed (Participants) | 39 | 38 | 27 | 30
  CD4 All Doubles - A/Indonesia, Month 18 | 2003.28 (964.77) | 1530.61 (1228.44) | 2975.66 (1696.72) | 2458.61 (1829.69)
  CD4 All Doubles - A/Vietnam, Month 18: number analyzed (Participants) | 42 | 43 | 30 | 32
  CD4 All Doubles - A/Vietnam, Month 18 | 2230.56 (1780.46) | 1628.90 (2059.72) | 2972.79 (1797.59) | 2535.97 (2627.53)
  CD4 CD40L - A/Vietnam, Day 0 | 536.99 (406.96) | 505.20 (497.95) | 504.23 (476.25) | 729.16 (736.68)
  CD4 CD40L - A/Vietnam, Month 6: number analyzed (Participants) | 32 | 31 | 36 | 28
  CD4 CD40L - A/Vietnam, Month 6 | 1272.27 (819.74) | 891.65 (657.93) | 1659.46 (823.79) | 1548.04 (918.09)
  CD4 CD40L - A/Indonesia, Month 12: number analyzed (Participants) | 33 | 34 | 23 | 31
  CD4 CD40L - A/Indonesia, Month 12 | 1361.91 (670.66) | 1209.07 (715.01) | 1610.40 (1079.91) | 1478.55 (1259.28)
  CD4 CD40L - A/Vietnam, Month 12: number analyzed (Participants) | 29 | 33 | 21 | 30
  CD4 CD40L - A/Vietnam, Month 12 | 1189.38 (519.31) | 1059.77 (917.49) | 1217.48 (1056.53) | 1173.39 (2904.15)
  CD4 CD40L - A/Indonesia, Month 12 + 7 Days: number analyzed (Participants) | 38 | 39 | 26 | 32
  CD4 CD40L - A/Indonesia, Month 12 + 7 Days | 1968.90 (1594.19) | 1724.77 (1242.19) | 2880.43 (1936.74) | 3101.88 (6940.95)
  CD4 CD40L - A/Vietnam, Month 12 + 7 Days: number analyzed (Participants) | 41 | 40 | 26 | 33
  CD4 CD40L - A/Vietnam, Month 12 + 7 Days | 2179.65 (2615.03) | 1781.72 (1287.53) | 2842.20 (2607.80) | 3365.20 (18999.95)
  CD4 CD40L - A/Indonesia, Month 12 + 21 Days: number analyzed (Participants) | 37 | 38 | 30 | 32
  CD4 CD40L - A/Indonesia, Month 12 + 21 Days | 2744.31 (1545.16) | 2097.74 (1860.85) | 3431.78 (2897.09) | 3124.45 (2787.90)
  CD4 CD40L - A/Vietnam, Month 12 + 21 Days: number analyzed (Participants) | 38 | 41 | 32 | 32
  CD4 CD40L - A/Vietnam, Month 12 + 21 Days | 2583.09 (2102.23) | 2184.58 (1371.47) | 3179.78 (3132.51) | 3479.95 (3622.29)
  CD4 CD40L - A/Indonesia, Month 18: number analyzed (Participants) | 39 | 38 | 27 | 30
  CD4 CD40L - A/Indonesia, Month 18 | 1943.30 (922.92) | 1532.05 (1186.69) | 2859.97 (1657.11) | 2317.11 (1865.51)
  CD4 CD40L - A/Vietnam, Month 18: number analyzed (Participants) | 42 | 43 | 30 | 32
  CD4 CD40L - A/Vietnam, Month 18 | 2174.81 (1734.47) | 1755.83 (1930.06) | 2849.08 (1755.65) | 2483.47 (2583.46)
  CD4 IL-2 - A/Vietnam, Day 0 | 376.07 (336.28) | 409.33 (480.49) | 436.65 (411.16) | 612.11 (632.55)
  CD4 IL-2 - A/Vietnam, Month 6: number analyzed (Participants) | 32 | 31 | 36 | 28
  CD4 IL-2 - A/Vietnam, Month 6 | 1097.97 (712.55) | 804.03 (632.15) | 1461.85 (769.17) | 1403.84 (915.32)
  CD4 IL-2 - A/Indonesia, Month 12: number analyzed (Participants) | 33 | 34 | 23 | 31
  CD4 IL-2 - A/Indonesia, Month 12 | 1149.50 (571.65) | 1065.33 (661.19) | 1517.94 (1028.90) | 1293.00 (1103.73)
  CD4 IL-2 - A/Vietnam, Month 12: number analyzed (Participants) | 29 | 33 | 21 | 30
  CD4 IL-2 - A/Vietnam, Month 12 | 992.70 (427.17) | 814.08 (714.13) | 1083.65 (1008.19) | 1048.97 (2636.29)
  CD4 IL-2 - A/Indonesia, Month 12 + 7 Days: number analyzed (Participants) | 38 | 39 | 26 | 32
  CD4 IL-2 - A/Indonesia, Month 12 + 7 Days | 1498.36 (1396.73) | 1476.33 (1015.37) | 2543.33 (1712.80) | 2670.96 (5571.66)
  CD4 IL-2 - A/Vietnam, Month 12 + 7 Days: number analyzed (Participants) | 41 | 40 | 26 | 33
  CD4 IL-2 - A/Vietnam, Month 12 + 7 Days | 1897.17 (2415.04) | 1533.21 (1397.88) | 2477.58 (2347.38) | 2942.81 (17299.39)
  CD4 IL-2 - A/Indonesia, Month 12 + 21 Days: number analyzed (Participants) | 37 | 38 | 30 | 32
  CD4 IL-2 - A/Indonesia, Month 12 + 21 Days | 2392.88 (1398.76) | 1858.04 (1721.69) | 3108.60 (2632.60) | 2747.73 (2516.72)
  CD4 IL-2 - A/Vietnam, Month 12 + 21 Days: number analyzed (Participants) | 38 | 41 | 32 | 32
  CD4 IL-2 - A/Vietnam, Month 12 + 21 Days | 2268.27 (1995.17) | 1932.19 (1276.22) | 2992.35 (2869.19) | 3105.21 (3366.65)
  CD4 IL-2 - A/Indonesia, Month 18: number analyzed (Participants) | 39 | 38 | 27 | 30
  CD4 IL-2 - A/Indonesia, Month 18 | 1703.60 (838.53) | 1383.29 (1077.39) | 2559.41 (1683.14) | 2104.29 (1607.98)
  CD4 IL-2 - A/Vietnam, Month 18: number analyzed (Participants) | 42 | 43 | 30 | 32
  CD4 IL-2 - A/Vietnam, Month 18 | 1869.31 (1525.68) | 1394.95 (1933.81) | 2589.97 (1776.18) | 2162.08 (2461.02)
  CD4 IFN-γ - A/Vietnam, Day 0 | 410.28 (363.50) | 336.74 (443.20) | 379.98 (364.14) | 476.66 (687.60)
  CD4 IFN-γ - A/Vietnam, Month 6: number analyzed (Participants) | 32 | 31 | 36 | 28
  CD4 IFN-γ - A/Vietnam, Month 6 | 690.45 (600.77) | 539.79 (432.94) | 771.40 (459.71) | 748.72 (758.34)
  CD4 IFN-γ - A/Indonesia, Month 12: number analyzed (Participants) | 33 | 34 | 23 | 31
  CD4 IFN-γ - A/Indonesia, Month 12 | 716.74 (400.83) | 609.84 (578.82) | 832.27 (746.45) | 794.44 (765.51)
  CD4 IFN-γ - A/Vietnam, Month 12: number analyzed (Participants) | 29 | 33 | 21 | 30
  CD4 IFN-γ - A/Vietnam, Month 12 | 729.77 (345.26) | 565.44 (574.28) | 633.07 (650.52) | 767.14 (1198.67)
  CD4 IFN-γ - A/Indonesia, Month 12 + 7 Days: number analyzed (Participants) | 38 | 39 | 26 | 32
  CD4 IFN-γ - A/Indonesia, Month 12 + 7 Days | 973.45 (756.29) | 812.11 (693.80) | 1308.07 (966.01) | 1560.86 (2907.99)
  CD4 IFN-γ - A/Vietnam, Month 12 + 7 Days: number analyzed (Participants) | 41 | 40 | 26 | 33
  CD4 IFN-γ - A/Vietnam, Month 12 + 7 Days | 1131.19 (1352.73) | 892.51 (905.48) | 1335.77 (1104.69) | 1635.21 (7167.21)
  CD4 IFN-γ - A/Indonesia, Month 12 + 21 Days: number analyzed (Participants) | 37 | 38 | 30 | 32
  CD4 IFN-γ - A/Indonesia, Month 12 + 21 Days | 1245.91 (936.91) | 948.13 (1366.34) | 1540.77 (1136.61) | 1662.38 (1310.77)
  CD4 IFN-γ - A/Vietnam, Month 12 + 21 Days: number analyzed (Participants) | 38 | 41 | 32 | 32
  CD4 IFN-γ - A/Vietnam, Month 12 + 21 Days | 1278.22 (1209.43) | 1074.61 (717.53) | 1539.76 (1287.82) | 1795.04 (2122.78)
  CD4 IFN-γ - A/Indonesia, Month 18: number analyzed (Participants) | 39 | 38 | 27 | 30
  CD4 IFN-γ - A/Indonesia, Month 18 | 1113.27 (598.27) | 902.31 (742.69) | 1329.00 (814.58) | 1292.88 (1081.31)
  CD4 IFN-γ - A/Vietnam, Month 18: number analyzed (Participants) | 42 | 43 | 30 | 32
  CD4 IFN-γ - A/Vietnam, Month 18 | 1309.65 (1177.92) | 901.99 (1416.15) | 1418.76 (1038.94) | 1284.53 (1281.98)
  CD4 TNF-α - A/Vietnam, Day 0 | 355.17 (302.08) | 287.10 (423.56) | 341.11 (356.99) | 512.64 (572.95)
  CD4 TNF-α - A/Vietnam, Month 6: number analyzed (Participants) | 32 | 31 | 36 | 28
  CD4 TNF-α - A/Vietnam, Month 6 | 886.97 (662.75) | 629.87 (556.20) | 1187.24 (710.18) | 1180.29 (829.76)
  CD4 TNF-α - A/Indonesia, Month 12: number analyzed (Participants) | 33 | 34 | 23 | 31
  CD4 TNF-α - A/Indonesia, Month 12 | 1020.53 (642.48) | 896.53 (690.42) | 1251.38 (970.03) | 995.80 (1066.30)
  CD4 TNF-α - A/Vietnam, Month 12: number analyzed (Participants) | 29 | 33 | 21 | 30
  CD4 TNF-α - A/Vietnam, Month 12 | 886.76 (457.39) | 673.80 (651.52) | 790.01 (938.28) | 903.64 (2220.85)
  CD4 TNF-α - A/Indonesia, Month 12 + 7 Days: number analyzed (Participants) | 38 | 39 | 26 | 32
  CD4 TNF-α - A/Indonesia, Month 12 + 7 Days | 1198.25 (1200.42) | 1217.50 (971.57) | 2108.88 (1380.62) | 2379.07 (5801.63)
  CD4 TNF-α - A/Vietnam, Month 12 + 7 Days: number analyzed (Participants) | 41 | 40 | 26 | 33
  CD4 TNF-α - A/Vietnam, Month 12 + 7 Days | 1289.39 (2162.71) | 1136.90 (1164.93) | 1997.48 (1725.20) | 2466.32 (16740.25)
  CD4 TNF-α - A/Indonesia, Month 12 + 21 Days: number analyzed (Participants) | 37 | 38 | 30 | 32
  CD4 TNF-α - A/Indonesia, Month 12 + 21 Days | 2047.96 (1439.33) | 1515.97 (1751.14) | 2800.66 (2480.69) | 2510.61 (2450.88)
  CD4 TNF-α - A/Vietnam, Month 12 + 21 Days: number analyzed (Participants) | 38 | 41 | 32 | 32
  CD4 TNF-α - A/Vietnam, Month 12 + 21 Days | 1833.81 (2015.18) | 1428.02 (1030.82) | 2373.80 (2542.38) | 2571.60 (3441.06)
  CD4 TNF-α - A/Indonesia, Month 18: number analyzed (Participants) | 39 | 38 | 27 | 30
  CD4 TNF-α - A/Indonesia, Month 18 | 1461.90 (863.23) | 1009.39 (1077.18) | 2445.88 (1505.10) | 1979.21 (1590.60)
  CD4 TNF-α - A/Vietnam, Month 18: number analyzed (Participants) | 42 | 43 | 30 | 32
  CD4 TNF-α - A/Vietnam, Month 18 | 1499.43 (1302.01) | 1250.85 (1843.92) | 2269.35 (1494.81) | 1914.16 (2270.93)
  CD8 All Doubles - A/Vietnam, Day 0: number analyzed (Participants) | 47 | 49 | 46 | 43
  CD8 All Doubles - A/Vietnam, Day 0 | 33.23 (473.07) | 30.79 (332.90) | 18.67 (297.54) | 21.71 (163.41)
  CD8 All Doubles - A/Vietnam, Month 6: number analyzed (Participants) | 32 | 31 | 36 | 28
  CD8 All Doubles - A/Vietnam, Month 6 | 56.22 (359.78) | 60.15 (348.65) | 31.83 (296.96) | 34.66 (208.62)
  CD8 All Doubles - A/Indonesia, Month 12: number analyzed (Participants) | 32 | 30 | 17 | 30
  CD8 All Doubles - A/Indonesia, Month 12 | 41.20 (285.40) | 19.96 (258.08) | 33.27 (237.99) | 34.16 (449.53)
  CD8 All Doubles - A/Vietnam, Month 12: number analyzed (Participants) | 28 | 28 | 17 | 27
  CD8 All Doubles - A/Vietnam, Month 12 | 14.72 (293.17) | 13.96 (149.10) | 8.90 (107.93) | 30.14 (365.90)
  CD8 All Doubles - A/Indonesia, Month 12 + 7 Days: number analyzed (Participants) | 34 | 31 | 22 | 26
  CD8 All Doubles - A/Indonesia, Month 12 + 7 Days | 68.32 (385.82) | 48.09 (292.33) | 41.66 (276.01) | 57.43 (369.42)
  CD8 All Doubles - A/Vietnam, Month 12 + 7 Days: number analyzed (Participants) | 31 | 33 | 23 | 25
  CD8 All Doubles - A/Vietnam, Month 12 + 7 Days | 18.73 (398.89) | 23.11 (409.70) | 9.04 (325.93) | 62.81 (426.34)
  CD8 All Doubles - A/Indonesia, Month 12 + 21 Days: number analyzed (Participants) | 34 | 37 | 27 | 31
  CD8 All Doubles - A/Indonesia, Month 12 + 21 Days | 59.21 (402.04) | 22.21 (196.85) | 42.28 (213.86) | 60.95 (301.71)
  CD8 All Doubles - A/Vietnam, Month 12 + 21 Days: number analyzed (Participants) | 38 | 39 | 28 | 31
  CD8 All Doubles - A/Vietnam, Month 12 + 21 Days | 16.35 (341.81) | 10.06 (260.79) | 16.58 (227.02) | 51.01 (320.71)
  CD8 All Doubles - A/Indonesia, Month 18: number analyzed (Participants) | 34 | 36 | 24 | 28
  CD8 All Doubles - A/Indonesia, Month 18 | 45.87 (268.24) | 36.98 (349.38) | 29.12 (194.72) | 36.73 (391.36)
  CD8 All Doubles - A/Vietnam, Month 18: number analyzed (Participants) | 41 | 39 | 28 | 29
  CD8 All Doubles - A/Vietnam, Month 18 | 27.14 (378.73) | 17.52 (231.65) | 26.49 (396.90) | 17.79 (189.35)
  CD8 CD40L - A/Vietnam, Day 0: number analyzed (Participants) | 47 | 49 | 46 | 43
  CD8 CD40L - A/Vietnam, Day 0 | 3.05 (54.73) | 3.22 (55.84) | 2.48 (130.89) | 2.79 (19.72)
  CD8 CD40L - A/Vietnam, Month 6: number analyzed (Participants) | 32 | 31 | 36 | 28
  CD8 CD40L - A/Vietnam, Month 6 | 2.59 (24.33) | 3.07 (55.80) | 3.00 (101.52) | 1.51 (20.14)
  CD8 CD40L - A/Indonesia, Month 12: number analyzed (Participants) | 32 | 30 | 17 | 30
  CD8 CD40L - A/Indonesia, Month 12 | 2.09 (28.38) | 3.66 (26.90) | 4.44 (40.48) | 4.48 (83.08)
  CD8 CD40L - A/Vietnam, Month 12: number analyzed (Participants) | 28 | 28 | 17 | 27
  CD8 CD40L - A/Vietnam, Month 12 | 2.33 (34.71) | 2.47 (32.62) | 2.16 (52.15) | 2.87 (40.66)
  CD8 CD40L - A/Indonesia, Month 12 + 7 Days: number analyzed (Participants) | 34 | 31 | 22 | 26
  CD8 CD40L - A/Indonesia, Month 12 + 7 Days | 8.21 (51.25) | 7.68 (119.95) | 13.23 (99.16) | 7.76 (99.48)
  CD8 CD40L - A/Vietnam, Month 12 + 7 Days: number analyzed (Participants) | 31 | 33 | 23 | 25
  CD8 CD40L - A/Vietnam, Month 12 + 7 Days | 4.40 (30.87) | 2.90 (183.17) | 2.90 (39.63) | 10.59 (52.19)
  CD8 CD40L - A/Indonesia, Month 12 + 21 Days: number analyzed (Participants) | 34 | 37 | 27 | 31
  CD8 CD40L - A/Indonesia, Month 12 + 21 Days | 5.43 (73.31) | 5.98 (61.91) | 8.29 (57.18) | 7.45 (96.27)
  CD8 CD40L - A/Vietnam, Month 12 + 21 Days: number analyzed (Participants) | 38 | 39 | 28 | 31
  CD8 CD40L - A/Vietnam, Month 12 + 21 Days | 3.96 (67.70) | 2.44 (92.98) | 3.11 (32.25) | 3.70 (34.54)
  CD8 CD40L - A/Indonesia, Month 18: number analyzed (Participants) | 34 | 36 | 24 | 28
  CD8 CD40L - A/Indonesia, Month 18 | 3.52 (49.19) | 4.22 (56.87) | 2.45 (37.14) | 2.75 (36.15)
  CD8 CD40L - A/Vietnam, Month 18: number analyzed (Participants) | 41 | 39 | 28 | 43
  CD8 CD40L - A/Vietnam, Month 18 | 4.32 (59.02) | 3.84 (75.59) | 4.78 (62.03) | 2.09 (59.01)
  CD8 IL-2 - A/Vietnam, Day 0: number analyzed (Participants) | 47 | 49 | 46 | 43
  CD8 IL-2 - A/Vietnam, Day 0 | 18.34 (169.79) | 22.25 (202.40) | 10.40 (167.00) | 15.03 (86.58)
  CD8 IL-2 - A/Vietnam, Month 6: number analyzed (Participants) | 32 | 31 | 36 | 28
  CD8 IL-2 - A/Vietnam, Month 6 | 24.13 (246.71) | 30.85 (186.03) | 16.53 (173.90) | 19.63 (145.48)
  CD8 IL-2 - A/Indonesia, Month 12: number analyzed (Participants) | 32 | 30 | 17 | 30
  CD8 IL-2 - A/Indonesia, Month 12 | 29.84 (250.29) | 18.29 (246.48) | 17.80 (236.04) | 28.56 (430.21)
  CD8 IL-2 - A/Vietnam, Month 12: number analyzed (Participants) | 28 | 28 | 17 | 27
  CD8 IL-2 - A/Vietnam, Month 12 | 9.12 (276.25) | 12.06 (148.06) | 8.22 (80.21) | 35.92 (362.09)
  CD8 IL-2 - A/Indonesia, Month 12 + 7 Days: number analyzed (Participants) | 34 | 31 | 22 | 26
  CD8 IL-2 - A/Indonesia, Month 12 + 7 Days | 55.96 (393.80) | 36.88 (268.94) | 28.07 (261.31) | 61.72 (318.59)
  CD8 IL-2 - A/Vietnam, Month 12 + 7 Days: number analyzed (Participants) | 31 | 33 | 23 | 25
  CD8 IL-2 - A/Vietnam, Month 12 + 7 Days | 20.48 (385.51) | 23.40 (399.09) | 8.29 (278.07) | 52.32 (392.40)
  CD8 IL-2 - A/Indonesia, Month 12 + 21 Days: number analyzed (Participants) | 34 | 37 | 27 | 31
  CD8 IL-2 - A/Indonesia, Month 12 + 21 Days | 62.99 (387.92) | 19.97 (198.10) | 31.51 (216.34) | 43.10 (277.22)
  CD8 IL-2 - A/Vietnam, Month 12 + 21 Days: number analyzed (Participants) | 38 | 39 | 28 | 31
  CD8 IL-2 - A/Vietnam, Month 12 + 21 Days | 12.52 (278.19) | 8.59 (207.18) | 14.20 (208.85) | 47.66 (280.88)
  CD8 IL-2 - A/Indonesia, Month 18: number analyzed (Participants) | 34 | 36 | 24 | 28
  CD8 IL-2 - A/Indonesia, Month 18 | 45.30 (266.64) | 31.29 (340.10) | 19.06 (157.42) | 31.56 (385.23)
  CD8 IL-2 - A/Vietnam, Month 18: number analyzed (Participants) | 41 | 39 | 28 | 29
  CD8 IL-2 - A/Vietnam, Month 18 | 15.35 (281.28) | 15.08 (211.25) | 14.48 (250.77) | 21.78 (153.80)
  CD8 IFN-γ - A/Vietnam, Day 0: number analyzed (Participants) | 47 | 49 | 46 | 43
  CD8 IFN-γ - A/Vietnam, Day 0 | 38.69 (468.52) | 22.01 (312.45) | 16.63 (273.01) | 24.90 (165.67)
  CD8 IFN-γ - A/Vietnam, Month 6: number analyzed (Participants) | 32 | 31 | 36 | 28
  CD8 IFN-γ - A/Vietnam, Month 6 | 31.09 (359.03) | 42.77 (334.23) | 24.28 (290.45) | 30.08 (200.12)
  CD8 IFN-γ - A/Indonesia, Month 12: number analyzed (Participants) | 32 | 30 | 17 | 30
  CD8 IFN-γ - A/Indonesia, Month 12 | 10.22 (195.65) | 6.58 (85.93) | 19.40 (172.59) | 13.70 (342.47)
  CD8 IFN-γ - A/Vietnam, Month 12: number analyzed (Participants) | 28 | 28 | 17 | 27
  CD8 IFN-γ - A/Vietnam, Month 12 | 5.79 (214.35) | 7.07 (174.18) | 4.31 (101.18) | 9.04 (120.34)
  CD8 IFN-γ - A/Indonesia, Month 12 + 7 Days: number analyzed (Participants) | 34 | 31 | 22 | 26
  CD8 IFN-γ - A/Indonesia, Month 12 + 7 Days | 13.38 (163.26) | 15.65 (111.26) | 10.25 (163.04) | 18.89 (170.88)
  CD8 IFN-γ - A/Vietnam, Month 12 + 7 Days: number analyzed (Participants) | 31 | 33 | 23 | 25
  CD8 IFN-γ - A/Vietnam, Month 12 + 7 Days | 7.58 (253.61) | 7.45 (181.01) | 7.59 (236.89) | 41.24 (348.65)
  CD8 IFN-γ - A/Indonesia, Month 12 + 21 Days: number analyzed (Participants) | 34 | 37 | 27 | 31
  CD8 IFN-γ - A/Indonesia, Month 12 + 21 Days | 13.88 (121.34) | 7.48 (123.95) | 6.66 (65.20) | 13.34 (135.85)
  CD8 IFN-γ - A/Vietnam, Month 12 + 21 Days: number analyzed (Participants) | 38 | 39 | 28 | 31
  CD8 IFN-γ - A/Vietnam, Month 12 + 21 Days | 11.90 (273.59) | 6.84 (235.75) | 6.18 (111.67) | 15.18 (269.18)
  CD8 IFN-γ - A/Indonesia, Month 18: number analyzed (Participants) | 34 | 36 | 24 | 28
  CD8 IFN-γ - A/Indonesia, Month 18 | 8.53 (121.12) | 12.19 (79.29) | 7.77 (113.83) | 6.53 (164.84)
  CD8 IFN-γ - A/Vietnam, Month 18: number analyzed (Participants) | 41 | 39 | 28 | 29
  CD8 IFN-γ - A/Vietnam, Month 18 | 13.33 (342.90) | 9.36 (182.90) | 5.10 (351.48) | 7.33 (135.83)
  CD8 TNF-α - A/Vietnam, Day 0: number analyzed (Participants) | 47 | 49 | 46 | 43
  CD8 TNF-α - A/Vietnam, Day 0 | 24.58 (437.31) | 19.36 (258.56) | 11.36 (179.18) | 14.50 (136.30)
  CD8 TNF-α - A/Vietnam, Month 6: number analyzed (Participants) | 32 | 31 | 36 | 28
  CD8 TNF-α - A/Vietnam, Month 6 | 31.78 (296.04) | 25.01 (272.87) | 26.33 (205.26) | 30.46 (172.62)
  CD8 TNF-α - A/Indonesia, Month 12: number analyzed (Participants) | 32 | 30 | 17 | 30
  CD8 TNF-α - A/Indonesia, Month 12 | 29.30 (263.60) | 15.38 (263.83) | 24.41 (194.37) | 25.59 (330.65)
  CD8 TNF-α - A/Vietnam, Month 12: number analyzed (Participants) | 28 | 28 | 17 | 27
  CD8 TNF-α - A/Vietnam, Month 12 | 8.92 (240.77) | 11.32 (106.95) | 6.46 (81.15) | 19.46 (337.02)
  CD8 TNF-α - A/Indonesia, Month 12 + 7 Days: number analyzed (Participants) | 34 | 31 | 22 | 26
  CD8 TNF-α - A/Indonesia, Month 12 + 7 Days | 54.30 (362.16) | 34.22 (261.37) | 35.18 (233.51) | 32.53 (309.18)
  CD8 TNF-α - A/Vietnam, Month 12 + 7 Days: number analyzed (Participants) | 31 | 33 | 23 | 25
  CD8 TNF-α - A/Vietnam, Month 12 + 7 Days | 10.89 (363.87) | 17.27 (340.50) | 8.21 (300.02) | 44.13 (394.01)
  CD8 TNF-α - A/Indonesia, Month 12 + 21 Days: number analyzed (Participants) | 34 | 37 | 27 | 31
  CD8 TNF-α - A/Indonesia, Month 12 + 21 Days | 48.83 (375.84) | 23.41 (155.91) | 31.57 (210.43) | 45.94 (281.82)
  CD8 TNF-α - A/Vietnam, Month 12 + 21 Days: number analyzed (Participants) | 38 | 39 | 28 | 31
  CD8 TNF-α - A/Vietnam, Month 12 + 21 Days | 14.75 (282.33) | 10.85 (228.98) | 8.45 (210.82) | 35.54 (288.39)
  CD8 TNF-α - A/Indonesia, Month 18: number analyzed (Participants) | 34 | 36 | 24 | 28
  CD8 TNF-α - A/Indonesia, Month 18 | 41.13 (261.84) | 24.97 (337.40) | 27.31 (164.07) | 31.10 (361.58)
  CD8 TNF-α - A/Vietnam, Month 18: number analyzed (Participants) | 41 | 39 | 28 | 29
  CD8 TNF-α - A/Vietnam, Month 18 | 16.41 (310.32) | 14.16 (217.05) | 16.70 (368.21) | 18.60 (170.85)

43. Secondary Outcome: GMTs of H5N1 Neutralizing Antibodies Against 2 Strains of Influenza Disease, for Adults Who Received Booster Dose at Month 6
Description: GMTs were calculated for H5N1 neutralizing antibodies against the A/Vietnam/1194/2004 or A/Indonesia/05/2005 strains.
Time Frame: At Day 0, Day 21, Day 42, Month 6, Month 6 + 7 Days, Month 6 + 21 Days and Month 12
Population: as for outcome 32
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 56 | 55 | 50 | 48
Titers
  A/Indonesia, Day 0 | 15.7 [14.5 to 17.0] | 15.5 [13.9 to 17.2] | 15.4 [14.1 to 16.9] | 14.4 [13.8 to 15.0]
  A/Indonesia, Day 21: number analyzed (Participants) | 56 | 55 | 7 | 11
  A/Indonesia, Day 21 | 39.8 [32.4 to 48.8] | 32.0 [26.6 to 38.5] | 37.9 [18.1 to 79.6] | 33.3 [19.1 to 58.2]
  A/Indonesia, Day 42: number analyzed (Participants) | 0 | 0 | 44 | 38
  A/Indonesia, Day 42 |  |  | 87.9 [68.1 to 113.4] | 75.9 [59.4 to 96.9]
  A/Indonesia, Month 6: number analyzed (Participants) | 55 | 49 | 49 | 48
  A/Indonesia, Month 6 | 22.0 [18.2 to 26.6] | 21.7 [18.1 to 25.9] | 41.7 [31.2 to 55.7] | 30.5 [23.7 to 39.3]
  A/Indonesia, Month 6 + 7 Days: number analyzed (Participants) | 53 | 47 | 48 | 46
  A/Indonesia, Month 6 + 7 Days | 966.7 [762.0 to 1226.3] | 512.4 [411.8 to 637.6] | 1016.1 [759.5 to 1359.4] | 562.0 [457.2 to 690.8]
  A/Indonesia, Month 6 + 21 Days: number analyzed (Participants) | 51 | 47 | 49 | 43
  A/Indonesia, Month 6 + 21 Days | 1815.5 [1368.0 to 2409.3] | 674.4 [536.9 to 847.1] | 2334.1 [1712.4 to 3181.4] | 831.3 [644.7 to 1071.8]
  A/Indonesia, Month 12: number analyzed (Participants) | 47 | 42 | 46 | 43
  A/Indonesia, Month 12 | 672.9 [527.4 to 858.7] | 392.1 [329.2 to 467.0] | 1003.8 [751.2 to 1341.4] | 540.0 [406.6 to 717.3]
  A/Vietnam, Day 0 | 20.4 [16.9 to 24.8] | 22.2 [17.8 to 27.6] | 18.9 [15.8 to 22.7] | 19.8 [16.2 to 24.1]
  A/Vietnam, Day 21: number analyzed (Participants) | 56 | 55 | 7 | 7
  A/Vietnam, Day 21 | 117.9 [91.8 to 151.5] | 106.7 [86.7 to 131.2] | 179.6 [93.5 to 345.0] | 78.8 [28.3 to 219.8]
  A/Vietnam, Day 42: number analyzed (Participants) | 0 | 0 | 44 | 41
  A/Vietnam, Day 42 |  |  | 372.3 [286.5 to 483.8] | 429.8 [319.1 to 578.9]
  A/Vietnam, Month 6: number analyzed (Participants) | 55 | 49 | 49 | 48
  A/Vietnam, Month 6 | 39.7 [30.8 to 51.0] | 39.2 [31.2 to 49.2] | 88.8 [64.0 to 123.1] | 91.2 [71.8 to 115.9]
  A/Vietnam, Month 6 + 7 Days: number analyzed (Participants) | 53 | 47 | 48 | 46
  A/Vietnam, Month 6 + 7 Days | 778.7 [623.8 to 972.1] | 1113.9 [857.8 to 1446.5] | 945.3 [729.8 to 1224.5] | 1058.8 [828.7 to 1352.8]
  A/Vietnam, Month 6 + 21 Days: number analyzed (Participants) | 52 | 47 | 49 | 45
  A/Vietnam, Month 6 + 21 Days | 1392.3 [1065.5 to 1819.2] | 1435.9 [1074.8 to 1918.4] | 1922.0 [1436.1 to 2572.4] | 1625.2 [1192.6 to 2214.6]
  A/Vietnam, Month 12: number analyzed (Participants) | 47 | 42 | 46 | 43
  A/Vietnam, Month 12 | 646.3 [539.0 to 775.0] | 762.9 [611.3 to 952.1] | 795.6 [577.1 to 1097.0] | 823.6 [600.5 to 1129.6]

44. Secondary Outcome: GMTs of H5N1 Neutralizing Antibodies Against 2 Strains of Influenza Disease, for Adults Who Received Booster Dose at Month 12
Description: GMTs were calculated for H5N1 neutralizing antibodies against the A/Vietnam/1194/2004 or A/Indonesia/05/2005 strains.
Time Frame: At Day 0, Day 21, Day 42, Month 6, Month 12, Month 12 + 7 Days and Month 12 + 21 Days
Population: as for outcome 32
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK1562902A V/I/12 Group | GSK1562902A V/V/12 Group | GSK1562902A 2V/I/12 Group | GSK1562902A 2V/V/12 Group
Number analyzed (Participants) | 59 | 60 | 55 | 55
Titers
  A/Indonesia, Day 0 | 15.8 [14.3 to 17.5] | 15.7 [14.4 to 17.2] | 15.1 [14.0 to 16.3] | 15.5 [14.1 to 17.0]
  A/Indonesia, Day 21: number analyzed (Participants) | 58 | 60 | 9 | 11
  A/Indonesia, Day 21 | 43.5 [35.0 to 54.0] | 37.0 [29.2 to 46.8] | 31.3 [18.3 to 53.5] | 26.5 [17.1 to 41.0]
  A/Indonesia, Day 42: number analyzed (Participants) | 0 | 0 | 48 | 48
  A/Indonesia, Day 42 |  |  | 97.0 [71.2 to 132.1] | 83.6 [67.8 to 103.0]
  A/Indonesia, Month 6: number analyzed (Participants) | 53 | 53 | 45 | 44
  A/Indonesia, Month 6 | 144.2 [107.2 to 194.0] | 122.4 [99.2 to 150.9] | 259.6 [195.6 to 344.5] | 196.3 [165.1 to 233.5]
  A/Indonesia, Month 12: number analyzed (Participants) | 52 | 51 | 44 | 41
  A/Indonesia, Month 12 | 124.7 [93.8 to 165.8] | 106.5 [80.2 to 141.5] | 234.6 [196.7 to 279.9] | 197.5 [155.0 to 251.6]
  A/Indonesia, Month 12 + 7 Days: number analyzed (Participants) | 51 | 49 | 42 | 40
  A/Indonesia, Month 12 + 7 Days | 2025.2 [1505.1 to 2725.1] | 936.9 [730.9 to 1200.9] | 2556.6 [1917.7 to 3408.4] | 1102.4 [770.2 to 1577.8]
  A/Indonesia, Month 12 + 21 Days: number analyzed (Participants) | 51 | 50 | 43 | 40
  A/Indonesia, Month 12 + 21 Days | 3254.2 [2325.5 to 4553.9] | 1301.5 [984.4 to 1720.7] | 4602.2 [3621.0 to 5849.3] | 1708.3 [1277.3 to 2284.8]
  A/Vietnam, Day 0: number analyzed (Participants) | 59 | 60 | 54 | 55
  A/Vietnam, Day 0 | 21.0 [17.2 to 25.5] | 20.6 [17.7 to 23.9] | 20.3 [16.7 to 24.6] | 20.0 [16.4 to 24.3]
  A/Vietnam, Day 21: number analyzed (Participants) | 58 | 60 | 8 | 9
  A/Vietnam, Day 21 | 124.4 [93.8 to 165.1] | 99.2 [80.2 to 122.6] | 80.2 [49.5 to 129.9] | 104.6 [35.3 to 310.0]
  A/Vietnam, Day 42: number analyzed (Participants) | 0 | 0 | 48 | 48
  A/Vietnam, Day 42 |  |  | 500.2 [360.5 to 693.9] | 404.4 [321.5 to 508.7]
  A/Vietnam, Month 6: number analyzed (Participants) | 53 | 53 | 45 | 45
  A/Vietnam, Month 6 | 270.6 [216.5 to 338.2] | 223.2 [191.7 to 259.9] | 401.9 [302.2 to 534.4] | 334.2 [267.0 to 418.3]
  A/Vietnam, Month 12: number analyzed (Participants) | 52 | 51 | 44 | 41
  A/Vietnam, Month 12 | 551.9 [431.3 to 706.4] | 504.0 [412.6 to 615.7] | 474.3 [395.3 to 568.9] | 468.1 [405.1 to 540.8]
  A/Vietnam, Month 12 + 7 Days: number analyzed (Participants) | 51 | 49 | 43 | 40
  A/Vietnam, Month 12 + 7 Days | 1848.1 [1453.8 to 2349.4] | 1448.5 [1175.5 to 1784.9] | 2002.2 [1533.7 to 2613.9] | 1718.1 [1301.3 to 2268.4]
  A/Vietnam, Month 12 + 21 Days: number analyzed (Participants) | 51 | 50 | 43 | 40
  A/Vietnam, Month 12 + 21 Days | 3209.7 [2461.3 to 4185.6] | 2520.3 [1914.2 to 3318.3] | 3874.7 [2944.6 to 5098.5] | 2304.8 [1747.6 to 3039.5]

45. Secondary Outcome: GMTs of H5N1 Neutralizing Antibodies Against 2 Strains of Influenza Disease, for Groups Who Received Booster Dose at Month 6
Description: GMTs were calculated for H5N1 neutralizing antibodies against the A/Vietnam/1194/2004 or A/Indonesia/05/2005 strains.
Time Frame: At Day 0, Day 21, Day 42, Month 6, Month 6 + 7 Days, Month 6 + 21 Days, Month 12 and Month 18
Population: The analysis was performed on the ATP Cohort for Persistence, which included all evaluable subjects for whom long term immunogenicity data were available and who complied with the inclusion/exclusion criteria as defined in the protocol. Day 42 data were available only from subjects who received 3 vaccine doses.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 51 | 49 | 47 | 44
Titers
  A/Indonesia, Day 0 | 15.7 [14.4 to 17.1] | 15.3 [13.7 to 17.1] | 15.5 [14.2 to 17.1] | 14.4 [13.8 to 15.1]
  A/Indonesia, Day 21: number analyzed (Participants) | 51 | 49 | 7 | 9
  A/Indonesia, Day 21 | 40.6 [32.5 to 50.6] | 31.8 [25.9 to 38.9] | 37.9 [18.1 to 79.6] | 36.4 [18.6 to 71.1]
  A/Indonesia, Day 42: number analyzed (Participants) | 0 | 0 | 41 | 36
  A/Indonesia, Day 42 |  |  | 86.3 [66.5 to 111.9] | 76.7 [61.0 to 96.3]
  A/Indonesia, Month 6: number analyzed (Participants) | 50 | 44 | 46 | 44
  A/Indonesia, Month 6 | 20.7 [17.4 to 24.7] | 22.2 [18.3 to 26.8] | 40.9 [30.3 to 55.0] | 29.2 [22.6 to 37.7]
  A/Indonesia, Month 6+ 7 Days: number analyzed (Participants) | 48 | 42 | 45 | 42
  A/Indonesia, Month 6+ 7 Days | 906.1 [708.4 to 1158.8] | 526.2 [419.4 to 660.2] | 963.3 [713.9 to 1299.9] | 537.3 [431.1 to 669.5]
  A/Indonesia, Month 6 + 21 Days: number analyzed (Participants) | 46 | 42 | 46 | 39
  A/Indonesia, Month 6 + 21 Days | 1703.0 [1263.7 to 2295.0] | 707.6 [556.5 to 899.8] | 2224.0 [1613.6 to 3065.3] | 814.7 [629.8 to 1053.8]
  A/Indonesia, Month 12: number analyzed (Participants) | 45 | 42 | 45 | 42
  A/Indonesia, Month 12 | 678.0 [525.5 to 874.7] | 392.1 [329.2 to 467.0] | 995.8 [740.6 to 1339.0] | 533.4 [399.2 to 712.8]
  A/Indonesia, Month 18: number analyzed (Participants) | 44 | 42 | 46 | 40
  A/Indonesia, Month 18 | 361.1 [283.8 to 459.6] | 225.0 [175.0 to 289.2] | 447.6 [345.2 to 580.5] | 290.1 [211.1 to 398.7]
  A/Vietnam, Day 0 | 20.9 [17.0 to 25.8] | 22.0 [17.5 to 27.6] | 19.3 [16.0 to 23.4] | 20.4 [16.5 to 25.2]
  A/Vietnam, Day 21: number analyzed (Participants) | 51 | 49 | 7 | 5
  A/Vietnam, Day 21 | 119.0 [91.5 to 154.7] | 109.0 [87.2 to 136.2] | 179.6 [93.5 to 345.0] | 103.6 [30.4 to 352.5]
  A/Vietnam, Day 42: number analyzed (Participants) | 0 | 0 | 41 | 39
  A/Vietnam, Day 42 |  |  | 352.9 [272.3 to 457.4] | 449.3 [338.8 to 596.0]
  A/Vietnam, Month 6: number analyzed (Participants) | 50 | 44 | 46 | 44
  A/Vietnam, Month 6 | 35.9 [28.2 to 45.6] | 39.8 [31.1 to 51.0] | 86.1 [61.6 to 120.4] | 91.4 [72.2 to 115.6]
  A/Vietnam, Month 6 + 7 Days: number analyzed (Participants) | 48 | 42 | 45 | 42
  A/Vietnam, Month 6 + 7 Days | 727.6 [579.8 to 913.0] | 1167.5 [893.0 to 1526.2] | 910.3 [700.4 to 1183.1] | 1035.0 [794.6 to 1348.1]
  A/Vietnam, Month 6 + 21 Days: number analyzed (Participants) | 47 | 42 | 46 | 41
  A/Vietnam, Month 6 + 21 Days | 1296.1 [985.1 to 1705.3] | 1568.2 [1176.0 to 2091.2] | 1863.6 [1387.9 to 2502.4] | 1609.1 [1162.2 to 2227.7]
  A/Vietnam, Month 12: number analyzed (Participants) | 45 | 42 | 45 | 42
  A/Vietnam, Month 12 | 643.3 [532.4 to 777.4] | 762.9 [611.3 to 952.1] | 797.7 [574.3 to 1107.9] | 844.7 [613.7 to 1162.7]
  A/Vietnam, Month 18: number analyzed (Participants) | 44 | 42 | 46 | 40
  A/Vietnam, Month 18 | 277.7 [208.2 to 370.3] | 338.1 [254.2 to 449.6] | 358.9 [254.4 to 506.2] | 444.5 [310.4 to 636.6]

46. Secondary Outcome: GMTs of H5N1 Neutralizing Antibodies Against 2 Strains of Influenza Disease, for Groups Who Received Booster Dose at Month 12
Description: GMTs were calculated for H5N1 neutralizing antibodies against the A/Vietnam/1194/2004 or A/Indonesia/05/2005 strains.
Time Frame: At Day 0, Day 21, Day 42, Month 6, Month 12, Month 12 + 7 Days, Month 12 + 21 Days and Month 18
Population: as for outcome 45
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A V/I/12 Group | GSK1562902A V/V/12 Group | GSK1562902A 2V/I/12 Group | GSK1562902A 2V/V/12 Group
Number analyzed (Participants) | 49 | 53 | 45 | 49
Titer
  A/Indonesia, Day 0 | 15.9 [14.2 to 17.9] | 15.6 [14.3 to 17.1] | 15.4 [14.0 to 16.9] | 15.7 [14.1 to 17.5]
  A/Indonesia, Day 21: number analyzed (Participants) | 49 | 53 | 9 | 10
  A/Indonesia, Day 21 | 45.1 [35.4 to 57.4] | 40.0 [31.1 to 51.5] | 31.3 [18.3 to 53.5] | 26.3 [16.1 to 43.0]
  A/Indonesia, Day 42: number analyzed (Participants) | 0 | 0 | 38 | 43
  A/Indonesia, Day 42 |  |  | 100.8 [68.6 to 148.1] | 80.7 [65.4 to 99.6]
  A/Indonesia, Month 6: number analyzed (Participants) | 49 | 51 | 42 | 44
  A/Indonesia, Month 6 | 146.5 [108.3 to 198.0] | 123.3 [99.6 to 152.6] | 255.0 [188.5 to 345.0] | 196.3 [165.1 to 233.5]
  A/Indonesia, Month 12: number analyzed (Participants) | 48 | 49 | 41 | 41
  A/Indonesia, Month 12 | 127.0 [95.7 to 168.5] | 107.8 [80.5 to 144.3] | 231.3 [191.6 to 279.3] | 197.5 [155.0 to 251.6]
  A/Indonesia, Month 12 + 7 Days: number analyzed (Participants) | 47 | 47 | 39 | 40
  A/Indonesia, Month 12 + 7 Days | 2190.6 [1657.3 to 2895.6] | 947.5 [732.7 to 1225.4] | 2476.1 [1839.2 to 3333.5] | 1102.4 [770.2 to 1577.8]
  A/Indonesia, Month 12 + 21 Days: number analyzed (Participants) | 47 | 48 | 40 | 40
  A/Indonesia, Month 12 + 21 Days | 3722.1 [2850.5 to 4860.1] | 1303.0 [975.7 to 1740.0] | 4661.0 [3625.1 to 5993.0] | 1708.3 [1277.3 to 2284.8]
  A/Indonesia, Month 18: number analyzed (Participants) | 45 | 49 | 39 | 40
  A/Indonesia, Month 18 | 903.0 [667.6 to 1221.5] | 423.7 [320.9 to 559.5] | 1708.9 [1243.6 to 2348.4] | 620.6 [475.5 to 809.9]
  A/Vietnam, Day 0: number analyzed (Participants) | 49 | 53 | 44 | 49
  A/Vietnam, Day 0 | 20.5 [16.5 to 25.4] | 20.8 [17.7 to 24.5] | 20.8 [16.6 to 26.1] | 20.5 [16.5 to 25.4]
  A/Vietnam, Day 21: number analyzed (Participants) | 49 | 53 | 8 | 8
  A/Vietnam, Day 21 | 123.7 [93.6 to 163.6] | 103.6 [82.1 to 130.8] | 80.2 [49.5 to 129.9] | 116.2 [33.9 to 398.1]
  A/Vietnam, Day 42: number analyzed (Participants) | 0 | 0 | 38 | 43
  A/Vietnam, Day 42 |  |  | 469.2 [321.4 to 684.8] | 399.2 [321.7 to 495.4]
  A/Vietnam, Month 6: number analyzed (Participants) | 49 | 51 | 42 | 45
  A/Vietnam, Month 6 | 274.5 [218.3 to 345.4] | 223.1 [190.4 to 261.4] | 405.1 [298.8 to 549.3] | 334.2 [267.0 to 418.3]
  A/Vietnam, Month 12: number analyzed (Participants) | 48 | 49 | 41 | 41
  A/Vietnam, Month 12 | 542.7 [417.6 to 705.2] | 511.2 [415.6 to 628.9] | 475.9 [393.1 to 576.1] | 468.1 [405.1 to 540.8]
  A/Vietnam, Month 12 + 7 Days: number analyzed (Participants) | 47 | 47 | 40 | 40
  A/Vietnam, Month 12 + 7 Days | 1945.3 [1532.8 to 2468.9] | 1435.4 [1163.3 to 1771.1] | 1972.2 [1490.9 to 2609.0] | 1718.1 [1301.3 to 2268.4]
  A/Vietnam, Month 12 + 21 Days: number analyzed (Participants) | 47 | 48 | 40 | 40
  A/Vietnam, Month 12 + 21 Days | 3490.4 [2712.8 to 4491.0] | 2495.4 [1886.4 to 3300.9] | 4057.4 [3048.1 to 5400.9] | 2304.8 [1747.6 to 3039.5]
  A/Vietnam, Month 18: number analyzed (Participants) | 44 | 48 | 39 | 40
  A/Vietnam, Month 18 | 813.2 [580.8 to 1138.5] | 585.9 [417.5 to 822.2] | 1650.0 [1203.4 to 2262.4] | 871.9 [621.0 to 1224.2]

47. Secondary Outcome: Number of Seroconverted Subjects for H5N1 Neutralizing Antibodies Against 2 Strains of Influenza Disease, for Groups Who Received Booster Dose at Month 6
Description: Seroconversion (SCR) was defined as the percentage of vaccinees with a minimum 4-fold increase in neutralizing antibody titer at the post-vaccination time-point compared to Day 0. The 2 flu strains assessed were A/Vietnam/1194/2004 (H5N1) and A/Indonesia/5/2005 (H5N1).
Time Frame: At Day 21, Day 42, Month 6, Month 6 + 7 Days, Month 6 + 21 Days and Month 12
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 56 | 55 | 49 | 48
Participants
  A/Indonesia, Day 21: number analyzed (Participants) | 56 | 55 | 7 | 11
  A/Indonesia, Day 21 | 19 | 13 | 1 | 4
  A/Indonesia, Day 42: number analyzed (Participants) | 0 | 0 | 44 | 38
  A/Indonesia, Day 42 |  |  | 32 | 28
  A/Indonesia, Month 6: number analyzed (Participants) | 55 | 49 | 49 | 48
  A/Indonesia, Month 6 | 6 | 5 | 20 | 13
  A/Indonesia, Month 6 + 7 Days: number analyzed (Participants) | 53 | 47 | 48 | 46
  A/Indonesia, Month 6 + 7 Days | 53 | 46 | 48 | 46
  A/Indonesia, Month 6 + 21 Days: number analyzed (Participants) | 51 | 47 | 49 | 43
  A/Indonesia, Month 6 + 21 Days | 51 | 47 | 49 | 43
  A/Indonesia, Month 12: number analyzed (Participants) | 47 | 42 | 46 | 43
  A/Indonesia, Month 12 | 47 | 42 | 46 | 42
  A/Vietnam, Day 21: number analyzed (Participants) | 56 | 55 | 7 | 7
  A/Vietnam, Day 21 | 40 | 34 | 5 | 5
  A/Vietnam, Day 42: number analyzed (Participants) | 0 | 0 | 44 | 41
  A/Vietnam, Day 42 |  |  | 42 | 39
  A/Vietnam, Month 6: number analyzed (Participants) | 55 | 49 | 49 | 48
  A/Vietnam, Month 6 | 18 | 10 | 28 | 31
  A/Vietnam, Month 6 + 7 Days: number analyzed (Participants) | 53 | 47 | 48 | 46
  A/Vietnam, Month 6 + 7 Days | 51 | 45 | 48 | 45
  A/Vietnam, Month 6 + 21 Days: number analyzed (Participants) | 52 | 47 | 49 | 45
  A/Vietnam, Month 6 + 21 Days | 52 | 45 | 49 | 45
  A/Vietnam, Month 12: number analyzed (Participants) | 47 | 42 | 46 | 43
  A/Vietnam, Month 12 | 47 | 42 | 45 | 42

48. Secondary Outcome: Number of Seroconverted Subjects for H5N1 Neutralizing Antibodies Against 2 Strains of Influenza Disease, for Groups Who Received Booster Dose at Month 12
Description: as for outcome 47
Time Frame: At Day 21, Day 42, Month 6, Month 12, Month 12 + 7 Days and Month 12 + 21 Days
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/12 Group | GSK1562902A V/V/12 Group | GSK1562902A 2V/I/12 Group | GSK1562902A 2V/V/12 Group
Number analyzed (Participants) | 58 | 60 | 48 | 48
Participants
  A/Indonesia, Day 21: number analyzed (Participants) | 58 | 60 | 9 | 11
  A/Indonesia, Day 21 | 19 | 17 | 1 | 1
  A/Indonesia, Day 42: number analyzed (Participants) | 0 | 0 | 48 | 48
  A/Indonesia, Day 42 |  |  | 35 | 32
  A/Indonesia, Month 6: number analyzed (Participants) | 53 | 53 | 45 | 44
  A/Indonesia, Month 6 | 45 | 44 | 43 | 44
  A/Indonesia, Month 12: number analyzed (Participants) | 52 | 51 | 44 | 41
  A/Indonesia, Month 12 | 41 | 39 | 42 | 40
  A/Indonesia, Month 12 + 7 Days: number analyzed (Participants) | 51 | 49 | 42 | 40
  A/Indonesia, Month 12 + 7 Days | 51 | 49 | 42 | 40
  A/Indonesia, Month 12 + 21 Days: number analyzed (Participants) | 51 | 50 | 43 | 40
  A/Indonesia, Month 12 + 21 Days | 50 | 50 | 43 | 40
  A/Vietnam, Day 21: number analyzed (Participants) | 58 | 60 | 8 | 9
  A/Vietnam, Day 21 | 40 | 38 | 4 | 5
  A/Vietnam, Day 42: number analyzed (Participants) | 0 | 0 | 47 | 48
  A/Vietnam, Day 42 |  |  | 43 | 45
  A/Vietnam, Month 6: number analyzed (Participants) | 53 | 53 | 44 | 45
  A/Vietnam, Month 6 | 51 | 50 | 40 | 41
  A/Vietnam, Month 12: number analyzed (Participants) | 52 | 51 | 43 | 41
  A/Vietnam, Month 12 | 48 | 49 | 43 | 40
  A/Vietnam, Month 12 + 7 Days: number analyzed (Participants) | 51 | 49 | 42 | 40
  A/Vietnam, Month 12 + 7 Days | 50 | 49 | 41 | 40
  A/Vietnam, Month 12 + 21 Days: number analyzed (Participants) | 51 | 50 | 42 | 40
  A/Vietnam, Month 12 + 21 Days | 51 | 50 | 42 | 39

49. Secondary Outcome: Number of Booster Seroconverted Subjects Against 2 Strains of Influenza Disease, for Groups Who Received Booster Dose at Month 6
Description: Booster SCR was defined as: For seronegative subjects at pre-booster (Month 6), antibody titer ≥ 1:40 at Month 6 + 7 days; For seropositive subjects at pre-booster (Month 6), antibody titer at Month 6 + 7 days ≥ 4 fold the pre-vaccination antibody titer at Month 6. The 2 flu strains assessed were A/Vietnam/1194/2004 and A/Indonesia/5/2005.
Time Frame: At Month 6 + 7 Days, Month 6 + 21 Days, Month 12 and Month 18
Population: This analysis was performed on the ATP Cohort for Immunogenicity (only for M12) and ATP Cohort for Persistence, which included all evaluable subjects for whom immunogenicity data/long term immunogenicity data were available and who complied with the inclusion/exclusion criteria as defined in the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group
Number analyzed (Participants) | 48 | 42 | 46 | 43
Participants
  A/Indonesia, Month 6 + 7 Days: number analyzed (Participants) | 48 | 42 | 45 | 42
  A/Indonesia, Month 6 + 7 Days | 48 | 41 | 43 | 41
  A/Indonesia, Month 6 + 21 Days: number analyzed (Participants) | 46 | 42 | 46 | 39
  A/Indonesia, Month 6 + 21 Days | 46 | 41 | 45 | 39
  A/Indonesia, Month 12: number analyzed (Participants) | 47 | 42 | 46 | 43
  A/Indonesia, Month 12 | 47 | 40 | 44 | 41
  A/Indonesia, Month 18: number analyzed (Participants) | 44 | 42 | 46 | 40
  A/Indonesia, Month 18 | 40 | 32 | 38 | 32
  A/Vietnam, Month 6 + 7 Days: number analyzed (Participants) | 48 | 42 | 45 | 43
  A/Vietnam, Month 6 + 7 Days | 44 | 40 | 35 | 38
  A/Vietnam, Month 6 + 21 Days: number analyzed (Participants) | 47 | 42 | 46 | 41
  A/Vietnam, Month 6 + 21 Days | 46 | 41 | 39 | 40
  A/Vietnam, Month 12: number analyzed (Participants) | 47 | 42 | 46 | 43
  A/Vietnam, Month 12 | 46 | 39 | 33 | 36
  A/Vietnam, Month 18: number analyzed (Participants) | 44 | 42 | 46 | 40
  A/Vietnam, Month 18 | 33 | 35 | 26 | 27

50. Secondary Outcome: Number of Booster Seroconverted Subjects Against 2 Strains of Influenza Disease, for Groups Who Received Booster Dose at Month 12
Description: Booster seroconversion (SCR) was defined as: For seronegative subjects at pre-booster (Month 12), antibody titer ≥ 1:40 at Month 12 + 7 days; For seropositive subjects at pre-booster (Month 12), antibody titer at Month 12 + 7 days ≥ 4 fold the pre-vaccination antibody titer at Month 12. The 2 flu strains assessed were A/Vietnam/1194/2004 and A/Indonesia/5/2005.
Time Frame: At Month 12 + 7 Days and Month 12 + 21 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/12 Group | GSK1562902A V/V/12 Group | GSK1562902A 2V/I/12 Group | GSK1562902A 2V/V/12 Group
Number analyzed (Participants) | 51 | 50 | 43 | 40
Participants
  A/Indonesia, Month 12 + 7 Days: number analyzed (Participants) | 51 | 49 | 42 | 40
  A/Indonesia, Month 12 + 7 Days | 42 | 35 | 34 | 20
  A/Indonesia, Month 12 + 21 Days | 46 | 39 | 42 | 29
  A/Vietnam, Month 12 + 7 Days: number analyzed (Participants) | 51 | 49 | 42 | 40
  A/Vietnam, Month 12 + 7 Days | 17 | 16 | 18 | 19
  A/Vietnam, Month 12 + 21 Days: number analyzed (Participants) | 51 | 50 | 42 | 40
  A/Vietnam, Month 12 + 21 Days | 31 | 25 | 31 | 21

51. Secondary Outcome: Number of Booster Seroconverted Subjects Against 2 Strains of Influenza Disease, for Groups Who Received Booster Dose at Month 12
Description: as for outcome 50
Time Frame: At Month 12 + 7 Days, Month 12 + 21 Days and Month 18
Population: as for outcome 40
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A V/I/12 Group | GSK1562902A V/V/12 Group | GSK1562902A 2V/I/12 Group | GSK1562902A 2V/V/12 Group
Number analyzed (Participants) | 47 | 48 | 40 | 40
Participants
  A/Indonesia, Month 12 + 7 Days: number analyzed (Participants) | 47 | 47 | 39 | 40
  A/Indonesia, Month 12 + 7 Days | 39 | 34 | 32 | 20
  A/Indonesia, Month 12 + 21 Days | 44 | 38 | 39 | 29
  A/Indonesia, Month 18: number analyzed (Participants) | 44 | 47 | 39 | 40
  A/Indonesia, Month 18 | 33 | 25 | 31 | 18
  A/Vietnam, Month 12 + 7 Days: number analyzed (Participants) | 47 | 47 | 39 | 40
  A/Vietnam, Month 12 + 7 Days | 15 | 15 | 17 | 19
  A/Vietnam, Month 12 + 21 Days: number analyzed (Participants) | 47 | 48 | 39 | 40
  A/Vietnam, Month 12 + 21 Days | 30 | 23 | 29 | 21
  A/Vietnam, Month 18: number analyzed (Participants) | 44 | 47 | 38 | 40
  A/Vietnam, Month 18 | 8 | 7 | 16 | 10

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicited AEs: during the 30-day (Days 0-29) post-primary and booster vaccination period; SAEs: during the entire study period (from Day 0 up to Month 18).
Arm/Group | GSK1562902A V/I/6 Group | GSK1562902A V/V/6 Group | GSK1562902A 2V/I/6 Group | GSK1562902A 2V/V/6 Group | GSK1562902A V/I/12 Group | GSK1562902A V/V/12 Group | GSK1562902A 2V/I/12 Group | GSK1562902A 2V/V/12 Group
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/66 | 0/64 | 0/63 | 0/64 | 1/64 | 0/65 | 0/63
Serious Adverse Events (participants affected / at risk) | 4/63 | 1/66 | 0/64 | 3/63 | 1/64 | 5/64 | 1/65 | 3/63
Other Adverse Events (participants affected / at risk) | 58/63 | 65/66 | 63/64 | 61/63 | 61/64 | 60/64 | 65/65 | 62/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1562902A V/I/6 Group (N=63) | GSK1562902A V/V/6 Group (N=66) | GSK1562902A 2V/I/6 Group (N=64) | GSK1562902A 2V/V/6 Group (N=63) | GSK1562902A V/I/12 Group (N=64) | GSK1562902A V/V/12 Group (N=64) | GSK1562902A 2V/I/12 Group (N=65) | GSK1562902A 2V/V/12 Group (N=63)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1562902A V/I/6 Group (N=63) | GSK1562902A V/V/6 Group (N=66) | GSK1562902A 2V/I/6 Group (N=64) | GSK1562902A 2V/V/6 Group (N=63) | GSK1562902A V/I/12 Group (N=64) | GSK1562902A V/V/12 Group (N=64) | GSK1562902A 2V/I/12 Group (N=65) | GSK1562902A 2V/V/12 Group (N=63)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (20) | 26 (34) | 27 (40) | 28 (47) | 20 (28) | 13 (21) | 29 (43) | 26 (35)
Chills (General disorders) | 22 (27) | 28 (33) | 24 (37) | 36 (53) | 22 (32) | 20 (24) | 25 (36) | 29 (49)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 4 (4)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 11 (13) | 8 (14) | 16 (24) | 13 (22) | 8 (10) | 11 (15) | 13 (21) | 15 (21)
Fatigue (General disorders) | 35 (48) | 37 (54) | 45 (84) | 44 (77) | 37 (57) | 33 (43) | 47 (75) | 44 (81)
Headache (Nervous system disorders) | 35 (47) | 34 (48) | 42 (78) | 42 (83) | 32 (48) | 34 (47) | 45 (76) | 41 (71)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 15 (16) | 18 (19) | 23 (34) | 20 (30) | 16 (18) | 7 (8) | 23 (29) | 25 (34)
Induration (General disorders) | 17 (22) | 13 (20) | 22 (35) | 25 (47) | 14 (18) | 16 (20) | 24 (38) | 19 (26)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 2 (3) | 3 (3) | 3 (4) | 0 (0) | 4 (4) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 41 (57) | 41 (61) | 48 (94) | 48 (92) | 49 (71) | 41 (60) | 45 (87) | 47 (88)
Nasopharyngitis (Infections and infestations) | 8 (10) | 5 (5) | 7 (7) | 11 (12) | 8 (8) | 8 (8) | 10 (11) | 5 (5)
Pain (General disorders) | 56 (96) | 62 (111) | 61 (157) | 59 (156) | 61 (107) | 57 (99) | 62 (154) | 58 (145)
Pyrexia (General disorders) | 6 (6) | 3 (4) | 4 (4) | 4 (4) | 5 (5) | 7 (8) | 5 (6) | 5 (6)
Swelling (General disorders) | 12 (14) | 15 (19) | 21 (32) | 22 (37) | 10 (11) | 13 (17) | 16 (22) | 16 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.